CLINICAL TRIAL: NCT02554812
Title: A PHASE 1B/2 OPEN-LABEL STUDY TO EVALUATE SAFETY, CLINICAL ACTIVITY, PHARMACOKINETICS AND PHARMACODYNAMICS OF AVELUMAB (MSB0010718C) IN COMBINATION WITH OTHER CANCER IMMUNOTHERAPIES IN PATIENTS WITH ADVANCED MALIGNANCIES
Brief Title: A Study Of Avelumab In Combination With Other Cancer Immunotherapies In Advanced Malignancies (JAVELIN Medley)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated since there was no need for further safety or efficacy data to be collected. The participants having benefit from the Investigational treatments have been moved to a continuation study (NCT05059522)
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: B9991004; 2015-002552-27 (EudraCT Number); JAVELIN MEDLEY (Other: Alias Study Number)
Record Dates: First submitted 2015-09-16; First posted 2015-09-18 (Estimated); Results first posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Advanced Cancer
Keywords: anti PD-L1; anti 4-1BB; OX40 agonist; anti M-CSF; TLR9 agonist; Non-small cell lung cancer (NSCLC); melanoma; squamous cell carcinoma of head and neck (SCCHN); triple negative breast cancer (TNBC); gastric cancer; Small cell lung cancer (SCLC); bladder cancer; platinum resistant ovarian cancer; TGCT/PVNS
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma; Squamous Cell Carcinoma of Head and Neck; Triple Negative Breast Neoplasms; Stomach Neoplasms; Small Cell Lung Carcinoma; Urinary Bladder Neoplasms | interventions — avelumab; utomilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (19):
- Cohort A1 (Experimental): NSCLC patients treated with avelumab + utomilumab (Dose level 1)
  Interventions: Drug: Avelumab; Drug: Utomilumab
- Cohort A2 (Experimental): NSCLC patients treated with avelumab + utomilumab (Dose level 2)
  Interventions: Drug: Avelumab; Drug: Utomilumab
- Cohort A3 (Experimental): NSCLC patients treated with avelumab + utomilumab (Dose level 3)
  Interventions: Drug: Avelumab; Drug: Utomilumab
- Cohort A4 (Experimental): Melanoma patients treated with avelumab +utomilumab
  Interventions: Drug: Avelumab; Drug: Utomilumab
- Cohort A5 (Experimental): SCCHN patients treated with avelumab + utomilumab
  Interventions: Drug: Avelumab; Drug: Utomilumab
- Cohort A6 (Experimental): TNBC patients treated with avelumab + utomilumab
  Interventions: Drug: Avelumab; Drug: Utomilumab
- Cohort A7 (Experimental): SCLC that has progressed after at least 1 line of platinum-containing therapy treated with avelumab +utomilumab
  Interventions: Drug: Avelumab; Drug: Utomilumab
- Cohort A8 (Experimental): NSCLC first-line Stage IV treated with avelumab +PF-05082566
  Interventions: Drug: Avelumab; Drug: Utomilumab
- Combination B Dose Escalation (Experimental): PF-04518600 + avelumab in selected tumor types
  Interventions: Drug: Avelumab; Drug: PF-04518600
- Combination B Expansion Cohorts (Experimental): PF-04518600 + avelumab in selected tumor types
  Interventions: Drug: Avelumab; Drug: PF-04518600
- Combination C Dose escalation cohorts (Experimental): PD 0360324 + avelumab in selected tumor types
  Interventions: Drug: Avelumab; Drug: PD 0360324
- Combination C Dose expansion cohorts (Experimental): PD 0360324 + aveluamb in selected tumor types
  Interventions: Drug: Avelumab; Drug: PD 0360324
- Combination D Dose escalation cohorts (Experimental): PF-05082566 + PF-04518600 + avelumab in selected tumor types
  Interventions: Drug: Avelumab; Drug: Utomilumab; Drug: PF-04518600
- Combination D Dose expansion cohorts (Experimental): PF-05082566 + PF-04518600 + avelumab in selected tumor types
  Interventions: Drug: Avelumab; Drug: Utomilumab; Drug: PF-04518600
- Cohort A9 (Experimental): NSCLC first-line Stage IV treated with avelumab +utomilumab (sequential starting with utomilumab monotherapy followed by combination)
  Interventions: Drug: Avelumab; Drug: Utomilumab
- Cohort A10 (Experimental): NSCLC first-line Stage IV treated with avelumab + utomilumab (sequential starting with avelumab monotherapy followed by combination)
  Interventions: Drug: Avelumab; Drug: Utomilumab
- Cohort F1 (Experimental): CMP-001 +avelumab in SCCHN
  Interventions: Drug: Avelumab; Drug: CMP-001
- Cohort F2 (Experimental): CMP-001+avelumab+utomilumab in SCCHN
  Interventions: Drug: Avelumab; Drug: Utomilumab; Drug: CMP-001
- Cohort F3 (Experimental): CMP-001 +avelumab+PF-04518600 in SCCHN
  Interventions: Drug: Avelumab; Drug: PF-04518600; Drug: CMP-001

INTERVENTIONS:
Drug: Avelumab — Anti-PD-L1 antibody
  Other Names: MSB0010718C
Drug: Utomilumab — Anti-4-1BB antibody
  Other Names: PF-05082566
  Arms: Cohort A1; Cohort A10; Cohort A2; Cohort A3; Cohort A4; Cohort A5; Cohort A6; Cohort A7; Cohort A8; Cohort A9; Cohort F2; Combination D Dose escalation cohorts; Combination D Dose expansion cohorts
Drug: PF-04518600 — OX40 Agonist
  Arms: Cohort F3; Combination B Dose Escalation; Combination B Expansion Cohorts; Combination D Dose escalation cohorts; Combination D Dose expansion cohorts
Drug: PD 0360324 — Anti-M-CSF
  Arms: Combination C Dose escalation cohorts; Combination C Dose expansion cohorts
Drug: CMP-001 — TLR9 agonist
  Arms: Cohort F1; Cohort F2; Cohort F3

SUMMARY:
This is a Phase 1b/2 dose-optimization study to evaluate safety, pharmacokinetics, pharmacodynamics, and preliminary antitumor activity of avelumab (MSB0010718C) in combination with other cancer immunotherapies in patients with locally advanced or metastatic solid tumors. The primary purpose is to assess the safety and early signs of efficacy of various avelumab combinations with other cancer immunotherapies, optimizing dosing regimens as appropriate, in a limited series of indications.

DETAILED DESCRIPTION:
This is a Phase 1b/2, open-label, multi-center, multiple-dose, safety, clinical activity, PK, and PD study of avelumab in combination with other immune modulators in adult patients with locally advanced or metastatic solid tumors (eg, non-small cell lung cancer (NSCLC), melanoma, squamous cell carcinoma of the head and neck (SCCHN), triple-negative breast cancer (TNBC), gastric cancer, platinum resistant ovarian cancer, bladder cancer, small cell lung cancer (SCLC) and progressing tenosynovial giant cell tumor/pigmented villonodular synovitis (TGCT/PVNS) . In Phase 1b, this includes patients whose disease has progressed on standard of care therapy or for whom no standard therapy is available. In Phase 2, enrollment criteria regarding prior treatment(s) received varies by tumor type. Incorporation of the other immune modulators into this study is based on preclinical and clinical data supportive of single-agent tolerability and potential clinical benefit, as well as non-clinical data suggesting safety, tolerability and clinical benefit of the agent(s) in combination with avelumab. Combinations of avelumab plus other immune modulator(s) to be evaluated are as follows:

* Combination A: avelumab plus utomilumab (4-1BB agonist mAb)
* Combination B: avelumab plus PF-04518600 (OX40 agonist mAb)
* Combination C: avelumab plus PD 0360324 (M-CSF mAb)
* Combination D: avelumab plus utomilumab plus PF-04518600
* Combination F: avelumab plus CMP-001 (TLR9 agonist) and avelumab plus CMP-001 plus utomilumab and avelumab plus CMP-001 and PF-04518600 Each combination will be studied individually in 2 study parts: 1) a Phase 1b Lead-in part to evaluate safety, and determine the maximum tolerated dose (MTD) or maximum administered dose (MAD) and RP2D (if applicable), of the combination, and 2) a Phase 2 part to evaluate efficacy and further evaluate safety of the selected dose from the Phase 1b portion in pre-specified patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of advanced/metastatic solid tumor. Measurable disease by RECIST 1.1 with at least 1 measurable lesion that has not been previously irradiated. Availability of tumor specimen taken within 1 year prior to study entry, with no intervening systemic anti-cancer therapy. No prior PD-1/PDL-1 therapy allowed. Combination A: Phase 1b, patients with NSCLC that have progressed on standard therapy or for which no standard therapy is available, and Phase 2, patients with NSCLC, melanoma, SCCHN, TNBC in any line of therapy, SCLC, 1st line NSCLC. 1st line NSCLC must demonstrate to express PD-L1. Activating EGFR mutation, ALK, ROS1 translocation/rearrangements are not permitted. Combination B: Phase 1b, patients with advanced solid tumors (NSCLC, SCCHN, melanoma) that have progressed on standard therapy or for which no standard therapy is available, and Phase 2, patients with NSCLC, melanoma, or SCCHN. Up to 2 lines of prior therapy in advanced/metastatic disease setting allowed. Activating EGFR mutation, ALK, ROS1 translocation/rearrangements are not permitted. Combination C: Ovarian cancer, SCCHN, NSCLC, gastric cancer, platinum resistant ovarian cancer. Up to 2 lines of prior therapy in advanced/metastatic disease setting allowed. TGCT/PVNS that is either inoperable or requires extensive resection. Prior treatment with agents targeting CSF-1/CSF-1R not allowed. NSCLC activating EGFR mutation, ALK, ROS1 translocation/rearrangements are not permitted. Combination D: NSCLC, melanoma, SCCHN, bladder cancer. NSCLC activating EGFR mutation, ALK, ROS1 translocation/rearrangements are not permitted. Up to 2 lines of prior therapy in advanced/metastatic disease setting allowed. Combination F: Recurrent or metastatic SCCHN. One to three prior lines of systemic therapy for advanced stage or metastatic disease. Patients must have received anti PD-1/PD-L1 containing therapy (requires at least two doses of PD-1/PD-L1 agent).Disease progression no earlier than 6 weeks from initiation of the latest anticancer therapy. Evidence of radiologic progression is required. • Patient must be a candidate for intralesional administration with at least one tumor lesion which can be injected safely.
* ECOG performance status 0 or 1
* Estimated life expectancy of at least 3 months
* Adequate bone marrow, renal, and liver function
* Resolved acute effects of prior therapy
* Negative serum pregnancy test at screening
* Male and female patients able to have children must agree to use at least 1 highly effective method of contraception throughout the study and for at least 90 days after last dose
* Signed and dated informed consent

Exclusion Criteria:

* Monoclonal antibody based anti-cancer therapy within 28 days prior to study entry or small-molecule based anti-cancer therapy (targeted therapy or chemotherapy) within 14 days prior to study entry. Combination F:PD-1/PD-L1 agent within 14 days prior study entry.
* Current or prior use of immunosuppressive medication within 7 days prior to study entry
* Active autoimmune disease requiring systemic steroids or immunosuppressive agents within 7 days prior to study entry
* Known prior or suspected hypersensitivity to investigational products
* Major surgery within 4 weeks or radiation therapy within 14 days prior to study entry
* Patients with known symptomatic brain metastases requiring steroids
* Previous high-dose chemotherapy requiring stem cell rescue
* Prior allogeneic stem cell transplant or organ graft
* Any of the following within 6 months prior to study entry: myocardial infarction, uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, or transient ischemic attack
* Symptomatic pulmonary embolism within 6 months prior to study entry
* Known HIV or AIDS-related illness
* Active infection requiring systemic therapy
* Positive HBV or HCV test indicating acute or chronic infection
* Administration of a live vaccine within 4 weeks prior to study entry
* Diagnosis of other malignancy within 5 years, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the breast or cervix, or low-grade (Gleason ≤6) prostate cancer
* Participation in other studies involving investigational drug(s) within 4 weeks prior to study entry and/or during study participation
* Persisting toxicity related to prior therapy >Grade 1
* Other severe acute or chronic medical condition
* Combo C :Existing periorbital edema.
* Combo C : Hypocalcemia, clinically significant bone disease or recent bone fracture (within 12 weeks prior study entry)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2015-11-09 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (87):
- United States (57):
  - UCSD Medical Center - Encinitas, Encinitas, California
  - Koman Family Outpatient Pavilion, La Jolla, California
  - UC San Diego Medical Center - La Jolla (Jacobs Medical Center / Thornton Pavilion), La Jolla, California
  - UC San Diego Perlman Medical Offices, La Jolla, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UCLA Clinical Research Unit (Adminstration Office), Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Hematology-Oncology Clinic, Los Angeles, California
  - UCLA Hematology-Oncology Infusion Center, Los Angeles, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - UCSD Medical Center - Vista, Vista, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Mount Sinai Comprehensive Cancer Center - Aventura, Aventura, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Michigan Hospitals, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Investigational Pharmacy, Karmanos Cancer Center, Detroit, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Karmanos Cancer Institute Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - VA NY Harbor Healthcare System, New York, New York
  - NYU Investigational Pharmacy, New York, New York
  - NYU Langone Medical Center, New York, New York
  - NYU Laura and Isaac Perlmutter Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Research Pharmacy #PH#, New York, New York
  - Weill Cornell Medical College/New York Presbyterian Hospital, New York, New York
  - Sampson Regional Medical Center, Clinton, North Carolina
  - Southeastern Medical Oncology Center, Clinton, North Carolina
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center, Jacksonville, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - UPCI Investigational Drug Service, Pittsburgh, Pennsylvania
  - UPMC Shadyside Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Sanford Cancer Center Oncology Clinic & Pharmacy, Sioux Falls, South Dakota
  - Sanford Gynecologic Oncology Clinic, Sioux Falls, South Dakota
  - Sanford Interventional Radiology, Sioux Falls, South Dakota
  - Sanford ENT Clinic, Sioux Falls, South Dakota
  - Sanford Research, Sioux Falls, South Dakota
  - Sanford USD Medical Center, Sioux Falls, South Dakota
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The Sarah Cannon Research Institute / Tennessee Oncology, PLLC, Nashville, Tennessee
  - Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - Vanderbilt University Oncology Pharmacy, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - UT Southwestern Simmons Comprehensive Cancer Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- Australia (12):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Macquarie University, Macquarie University, New South Wales
  - Melanoma Institute Australia, North Sydney, New South Wales
  - The Mater Hospital, North Sydney, New South Wales
  - Baxter Healthcare, Old Toongabie, New South Wales
  - Brighton Medical Imaging, Brighton, Victoria
  - Cabrini Hospital Brighton, Brighton, Victoria
  - Austin Health, Heidelberg, Victoria
  - Cabrini Hospital Malvern, Malvern, Victoria
  - Cabrini Hospital, Malvern, Victoria
  - Malvern Medical Imaging, Malvern, Victoria
  - Macquarie Heart, New South Wales
- Canada (6):
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - PH 145294, Centre Hospitalier de l'Universite de Montreal (CHUM), Oncology Research Pharmacy, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
- France (2):
  - Institut Gustave Roussy, Villejuif, Cedex
  - Institut Gustave Roussy, Villejuif
- Japan (2):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Cancer Center Hospital, Chuo-ku, Tokyo
- Poland (2):
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy, Warsaw, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy, Warsaw
- Taiwan (2):
  - Investigational Drug Services, National Taiwan University Hospital, Taipei
  - National Taiwan University Hospital, Taipei
- United Kingdom (4):
  - The Royal Marsden Hospital, London
  - The Royal Marsden NHS Foundation Trust, London
  - Sarah Cannon Research Institute UK, London
  - The Harley Street Clinic, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B9991004&StudyName=A%20Phase%201b%2F2%20Open-label%20Study%20To%20Evaluate%20Safety%2C%20Clinical%20Activity%2C%20Pharmacokinetics%20And%20Pharmacodynamics%20Of%20Avelumab%2A%20%28msb0010718c%29%20In%20Combination%20With%20Other%20Cancer%20Immunotherapies%20In%20Patients%20With%20Advanced%20Malignancies

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this study participants were evaluated in 5 different combinations with avelumab: Combination A, B, C, D and F. Each combination was planned to be conducted in 2 phases: Phase 1b (lead-in phase) and Phase 2 (expansion phase). Phase 2 was conducted at the selected dose level of avelumab combination which was determined safe for participants in Phase 1b.
Groups:
- Combination A Phase 1b NSCLC: Utomilumab 500 mg + Avelumab: During phase 1b participants with Non-Small Cell Lung Cancer (NSCLC) received utomilumab 500 mg intravenously (IV) every 4 weeks (Q4W) with 10 milligrams per kilogram (mg/kg) of avelumab administered IV every 2 weeks (Q2W) for 2 cycles, where each cycle was of 4 weeks.
- Combination A Phase 1b NSCLC: Utomilumab 100 mg + Avelumab: During phase 1b participants with NSCLC received utomilumab 100 mg IV Q4W with 10 mg/kg of avelumab administered IV Q2W for 2 cycles, where each cycle was of 4 weeks.
- Combination A Phase 1b NSCLC: Utomilumab 20 mg + Avelumab: During phase 1b participants with NSCLC received utomilumab 20 mg IV Q4W with 10 mg/kg of avelumab administered IV Q2W for 2 cycles, where each cycle was of 4 weeks.
- Combination A Phase 2 Melanoma: Utomilumab 100 mg + Avelumab: During Phase 2 participants with melanoma received utomilumab 100 mg IV Q4W with 10 mg/kg of avelumab administered IV Q2W for 2 cycles, where each cycle was of 4 weeks.
- Combination A Phase 2 SCCHN: Utomilumab 100 mg + Avelumab: During Phase 2 participants with Squamous Cell Carcinoma of the Head and Neck (SCCHN) received utomilumab 100 mg IV Q4W with 10 mg/kg of avelumab administered IV Q2W for 2 cycles, where each cycle was of 4 weeks.
- Combination A Phase 2 TNBC: Utomilumab 100 mg + Avelumab: During Phase 2 participants with Triple Negative Breast Cancer (TNBC) received utomilumab 100 mg IV Q4W with 10 mg/kg of avelumab administered IV Q2W for 2 cycles, where each cycle was of 4 weeks.
- Combination A Phase 2 SCLC: Utomilumab 100 mg + Avelumab: During Phase 2 participants with Squamous cell lung cancer (SCLC) received utomilumab 100 mg IV Q4W with 10 mg/kg of avelumab administered IV Q2W for 2 cycles, where each cycle was of 4 weeks.
- Combination A Phase 2 First Line (1L) NSCLC: Utomilumab 100 mg + Avelumab: During Phase 2 participants with NSCLC received utomilumab 100 mg IV Q4W with 10 mg/kg of avelumab administered IV Q2W for 2 cycles, where each cycle was of 4 weeks.
- Combination A Phase 2 1L NSCLC: Utomilumab Then Utomilumab + Avelumab: During Phase 2 participants with NSCLC received utomilumab 100 mg IV Q4W for cycle 1 then utomilumab 100 mg IV Q4W with 10 mg/kg of avelumab administered IV Q2W starting at cycle 2.
- Combination A Phase 2 1L NSCLC: Avelumab Then Utomilumab + Avelumab: During Phase 2 participants with NSCLC received avelumab 10 mg/kg administered IV Q2W for cycles 1 then utomilumab 100 mg IV Q4W with 10 mg/kg of avelumab administered IV Q2W starting at cycle 2.
- Combination B Phase 1b: PF-04518600 0.3 mg/kg + Avelumab: During Phase 1b participants received PF-04518600 0.3 mg/kg IV Q2W with 10 mg/kg of avelumab administered IV Q2W. Phase 2 in the melanoma cohort was not planned.
- Combination B Phase 1b: PF-04518600 1.0 mg/kg + Avelumab: During Phase 1b participants received PF-04518600 1.0 mg/kg IV Q2W with 10 mg/kg of avelumab administered IV Q2W. Phase 2 in the melanoma cohort was not planned.
- Combination B Phase 1b: PF-04518600 3.0 mg/kg + Avelumab: During Phase 1b participants received PF-04518600 3.0 mg/kg IV Q2W with 10 mg/kg of avelumab administered IV Q2W. Phase 2 in the melanoma cohort was not planned.
- Combination B Phase 2 NSCLC: PF-04518600 0.3 mg/kg + Avelumab: During Phase 2 participants with NSCLC received PF-04518600 0.3 mg/kg IV Q2W with 10 mg/kg of avelumab administered IV Q2W.
- Combination B Phase 2 SCCHN: PF-04518600 0.3 mg/kg + Avelumab: During Phase 2 participants with SCCHN received PF-04518600 0.3 mg/kg IV Q2W with 10 mg/kg of avelumab administered IV Q2W.
- Combination C Phase 1b: PD 0360324 50 mg + Avelumab: During Phase 1b participants received PD 0360324 50 mg IV Q2W with 10 mg/kg of avelumab administered IV Q2W for 2 cycles, where each cycle was of 4 weeks. Phase 2 was not planned.
- Combination C Phase 1b: PD 0360324 100 mg + Avelumab: During Phase 1b participants received PD 0360324 100 mg IV Q2W with 10 mg/kg of avelumab administered IV Q2W for 2 cycles, where each cycle was of 4 weeks.
- Combination C Phase 1b: PD 0360324 150 mg + Avelumab: During Phase 1b participants received PD 0360324 150 mg IV Q2W with 10 mg/kg of avelumab administered IV Q2W for 2 cycles, where each cycle was of 4 weeks.
- Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.1 mg/kg + Avelumab: During Phase 1b participants received utomilumab 20 mg IV Q4W along with PF-04518600 0.1 mg/kg IV Q2W and 10 mg/kg of avelumab administered IV Q2W for 2 cycles, where each cycle was of 4 weeks. Phase 2 was not planned.
- Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.1 mg/kg + Avelumab: During Phase 1b participants received utomilumab 50 mg IV Q4W along with PF-04518600 0.1 mg/kg IV Q2W and 10 mg/kg of avelumab administered IV Q2W for 2 cycles, where each cycle was of 4 weeks. Phase 2 was not planned.
- Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.3 mg/kg + Avelumab: During Phase 1b participants received utomilumab 20 mg IV Q4W along with PF-04518600 0.3 mg/kg IV Q2W and 10 mg/kg of avelumab administered IV Q2W for 2 cycles, where each cycle was of 4 weeks. Phase 2 was not planned.
- Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.3 mg/kg + Avelumab: During Phase 1b participants received utomilumab 50 mg IV Q4W along with PF-04518600 0.3 mg/kg IV Q2W and 10 mg/kg of avelumab administered IV Q2W for 2 cycles, where each cycle was of 4 weeks. Phase 2 was not planned.
- Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 1.0 mg/kg + Avelumab: During Phase 1b participants received utomilumab 20 mg IV Q4W along with PF-04518600 1.0 mg/kg IV Q2W and 10 mg/kg of avelumab administered IV Q2W for 2 cycles, where each cycle was of 4 weeks. Phase 2 was not planned.
- Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 1.0 mg/kg + Avelumab: During Phase 1b participants received utomilumab 50 mg IV Q4W along with PF-04518600 1.0 mg/kg IV Q2W and 10 mg/kg of avelumab administered IV Q2W for 2 cycles, where each cycle was of 4 weeks. Phase 2 was not planned.
- Combination F Phase 1b SCCHN: CMP-001 10 mg + Avelumab: During Phase 1b participants with SCCHN received CMP-001 at 10 mg for an initial 7 doses (2 sub-cutaneous [SC] administered at weekly intervals, followed by 5 intra tumoral [IT] administered at weekly intervals) and then administered IT Q2W for all cohorts along with 10 mg/kg of avelumab administered IV Q2W. Phase 2 was not planned.
- Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + Utomilumab 100 mg: During Phase 1b participants with SCCHN received CMP-001 at 10 mg for an initial 7 doses (2 SC administered at weekly intervals, followed by 5 IT administered at weekly intervals) and then administered IT Q2W for all cohorts along with 10 mg/kg of avelumab administered IV Q2W all cohorts plus utomilumab 100 mg administered IV Q4W. Phase 2 was not planned.
- Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + PF-04518600 0.3 mg/kg: During Phase 1b participants with SCCHN received CMP-001 at 10 mg for an initial 7 doses (2 SC administered at weekly intervals, followed by 5 IT administered at weekly intervals) and then administered IT Q2W for all cohorts along with 10 mg/kg of avelumab administered IV Q2W all cohorts plus PF-04518600 at 0.3 mg/kg administered IV Q2W. Phase 2 was not planned.
Period: Overall Study
Arm/Group | Combination A Phase 1b NSCLC: Utomilumab 500 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 20 mg + Avelumab | Combination A Phase 2 Melanoma: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCCHN: Utomilumab 100 mg + Avelumab | Combination A Phase 2 TNBC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 First Line (1L) NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 1L NSCLC: Utomilumab Then Utomilumab + Avelumab | Combination A Phase 2 1L NSCLC: Avelumab Then Utomilumab + Avelumab | Combination B Phase 1b: PF-04518600 0.3 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 1.0 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 3.0 mg/kg + Avelumab | Combination B Phase 2 NSCLC: PF-04518600 0.3 mg/kg + Avelumab | Combination B Phase 2 SCCHN: PF-04518600 0.3 mg/kg + Avelumab | Combination C Phase 1b: PD 0360324 50 mg + Avelumab | Combination C Phase 1b: PD 0360324 100 mg + Avelumab | Combination C Phase 1b: PD 0360324 150 mg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 1.0 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 1.0 mg/kg + Avelumab | Combination F Phase 1b SCCHN: CMP-001 10 mg + Avelumab | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + Utomilumab 100 mg | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + PF-04518600 0.3 mg/kg
Started | 29 | 28 | 29 | 28 | 35 | 21 | 10 | 21 | 11 | 11 | 12 | 12 | 8 | 14 | 25 | 10 | 8 | 6 | 12 | 12 | 12 | 12 | 12 | 11 | 6 | 7 | 7
Treated | 29 | 27 | 29 | 28 | 35 | 21 | 10 | 21 | 11 | 11 | 12 | 12 | 8 | 14 | 25 | 10 | 8 | 6 | 12 | 12 | 12 | 12 | 12 | 11 | 6 | 7 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 29 | 28 | 29 | 28 | 35 | 21 | 10 | 21 | 11 | 11 | 12 | 12 | 8 | 14 | 25 | 10 | 8 | 6 | 12 | 12 | 12 | 12 | 12 | 11 | 6 | 7 | 7
Not completed — Adverse Event | 2 | 5 | 3 | 0 | 5 | 0 | 1 | 6 | 2 | 2 | 1 | 2 | 0 | 3 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 2 | 1
Not completed — Death | 1 | 2 | 2 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Global deterioration of health status | 4 | 3 | 3 | 2 | 5 | 0 | 2 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 20 | 16 | 19 | 18 | 21 | 15 | 6 | 13 | 6 | 6 | 8 | 8 | 6 | 10 | 20 | 6 | 3 | 3 | 11 | 7 | 11 | 6 | 9 | 9 | 4 | 5 | 5
Not completed — Other | 0 | 0 | 2 | 3 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 2 | 2 | 3 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 3 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — No longer meets eligibility criteria | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination A Phase 1b NSCLC: Utomilumab 500 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 20 mg + Avelumab | Combination A Phase 2 Melanoma: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCCHN: Utomilumab 100 mg + Avelumab | Combination A Phase 2 TNBC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 First Line (1L) NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 1L NSCLC: Utomilumab Then Utomilumab + Avelumab | Combination A Phase 2 1L NSCLC: Avelumab Then Utomilumab + Avelumab | Combination B Phase 1b: PF-04518600 0.3 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 1.0 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 3.0 mg/kg + Avelumab | Combination B Phase 2 NSCLC: PF-04518600 0.3 mg/kg + Avelumab | Combination B Phase 2 SCCHN: PF-04518600 0.3 mg/kg + Avelumab | Combination C Phase 1b: PD 0360324 50 mg + Avelumab | Combination C Phase 1b: PD 0360324 100 mg + Avelumab | Combination C Phase 1b: PD 0360324 150 mg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 1.0 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 1.0 mg/kg + Avelumab | Combination F Phase 1b SCCHN: CMP-001 10 mg + Avelumab | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + Utomilumab 100 mg | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + PF-04518600 0.3 mg/kg | Total
Number analyzed (Participants) | 29 | 27 | 29 | 28 | 35 | 21 | 10 | 21 | 11 | 11 | 12 | 12 | 8 | 14 | 25 | 10 | 8 | 6 | 12 | 12 | 12 | 12 | 12 | 11 | 6 | 7 | 7 | 408
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.14 (11.22) | 60.74 (10.85) | 61.52 (11.81) | 63.71 (10.82) | 61.09 (11.80) | 53.33 (14.59) | 59.40 (12.74) | 65.24 (11.05) | 65.27 (10.05) | 69.55 (4.06) | 54.17 (12.55) | 64.75 (10.68) | 65.25 (10.39) | 66.64 (7.15) | 63.04 (8.12) | 62.50 (12.57) | 56.63 (9.32) | 54.33 (14.60) | 65.67 (10.65) | 63.50 (10.89) | 66.67 (10.29) | 61.58 (6.56) | 59.08 (11.29) | 61.36 (10.54) | 58.50 (16.29) | 66.14 (5.27) | 60.00 (21.63) | 62.11 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 15 | 8 | 4 | 21 | 4 | 9 | 5 | 7 | 5 | 7 | 3 | 9 | 3 | 7 | 3 | 1 | 3 | 3 | 6 | 3 | 3 | 1 | 1 | 0 | 0 | 149
  Male | 21 | 17 | 14 | 20 | 31 | 0 | 6 | 12 | 6 | 4 | 7 | 5 | 5 | 5 | 22 | 3 | 5 | 5 | 9 | 9 | 6 | 9 | 9 | 10 | 5 | 7 | 7 | 259
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 2 | 1 | 0 | 2 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 18
  Not Hispanic or Latino | 26 | 26 | 27 | 26 | 32 | 19 | 8 | 19 | 11 | 11 | 11 | 11 | 7 | 13 | 25 | 9 | 6 | 6 | 9 | 10 | 11 | 12 | 12 | 11 | 5 | 6 | 7 | 376
  Unknown or Not Reported | 2 | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 5 | 5 | 7 | 1 | 4 | 3 | 0 | 1 | 3 | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 3 | 2 | 4 | 1 | 0 | 0 | 0 | 0 | 46
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 3 | 1 | 0 | 2 | 6 | 0 | 2 | 1 | 1 | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 30
  White | 22 | 19 | 21 | 26 | 25 | 10 | 8 | 16 | 6 | 8 | 9 | 8 | 6 | 10 | 23 | 9 | 7 | 4 | 7 | 8 | 10 | 7 | 11 | 11 | 5 | 5 | 4 | 305
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 1 | 3 | 2 | 1 | 2 | 1 | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 25

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b Lead-in: Number of Participants With First 2 Cycles Dose Limiting Toxicity (DLT) for Combination A
Description: Severity of AEs graded as per CTCAE v4.03. Phase 1b lead-in, AEs occurring during DLT observation period, that attributable to one or more study drug in combination was classified as DLT: Hematologic: Grade (G)4 neutropenia lasting >7 day; Febrile neutropenia; Neutropenic infection; G >=3 thrombocytopenia with bleeding; G4 thrombocytopenia; G4 anemia. Non-Hematologic (Non-Laboratory): Any G3 toxicity, except following: Transient (24 H) G3 fatigue, local reaction, or headache that resolved to G1; G3-4 nausea/vomiting controlled by medical therapy within 72H; G3 hypertension controlled by medical therapy; G3 diarrhea improved to G <=2 within 72H after medical therapy; G3 skin toxicity resolved to G <=1 in <7 days after medical management; G >=3 amylase or lipase abnormality not associated with pancreatitis;G3 endocrinopathies controlled with medical therapy; Tumor flare phenomenon.G4 or G3 CRS lasting >24 H despite treatment.
Time Frame: Baseline up to Cycle 2 (up to 8 weeks)
Population: The analysis population included all participants enrolled in Phase 1b who were in the safety analysis set (all participants who received at least one dose of study drug) and received at least 75% of the prescribed doses unless due to treatment-related toxicity or either experienced DLT during the first 2 cycles (1 cycle = 4 weeks) or completed observation period for the first 2 cycles of treatment. Here, "N''=number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination A Phase 1b NSCLC: Utomilumab 500 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 20 mg + Avelumab
Number analyzed (Participants) | 29 | 28 | 29
Participants | 0 | 0 | 0

2. Primary Outcome: Phase 1b Lead-in: Number of Participants With First 2 Cycles DLT for Combination B
Description: as for outcome 1
Time Frame: Baseline up to Cycle 2 (up to 8 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combination B Phase 1b: PF-04518600 0.3 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 1.0 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 3.0 mg/kg + Avelumab
Number analyzed (Participants) | 12 | 12 | 8
Participants | 0 | 0 | 0

3. Primary Outcome: Phase 1b Lead-in: Number of Participants With First 2 Cycles DLT for Combination C
Description: as for outcome 1
Time Frame: Baseline up to Cycle 2 (up to 8 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combination C Phase 1b: PD 0360324 50 mg + Avelumab | Combination C Phase 1b: PD 0360324 100 mg + Avelumab | Combination C Phase 1b: PD 0360324 150 mg + Avelumab
Number analyzed (Participants) | 10 | 8 | 6
Participants | 0 | 0 | 0

4. Primary Outcome: Phase 1b Lead-in: Number of Participants With First 2 Cycles DLT for Combination D
Description: as for outcome 1
Time Frame: Baseline up to Cycle 2 (up to 8 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 1.0 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 1.0 mg/kg + Avelumab
Number analyzed (Participants) | 11 | 10 | 11 | 9 | 11 | 8
Participants | 1 | 0 | 0 | 2 | 1 | 0

5. Primary Outcome: Phase 1b Lead-in: Number of Participants With First Cycle DLT for Combination F
Description: as for outcome 1
Time Frame: Baseline up to first Cycle (up to 4 weeks)
Population: The analysis population included all participants enrolled in Phase 1b who were in the safety analysis set (all participants who received at least one dose of study drug) and received at least 75% of the prescribed doses unless due to treatment-related toxicity or either experienced DLT during the first cycle (1 cycle = 4 weeks) or completed observation period for the first cycle of treatment. Here, "N''=number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination F Phase 1b SCCHN: CMP-001 10 mg + Avelumab | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + Utomilumab 100 mg | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + PF-04518600 0.3 mg/kg
Number analyzed (Participants) | 6 | 6 | 6
Participants | 1 | 1 | 0

6. Primary Outcome: Phase 2: Percentage of Participants With Confirmed Objective Response (OR) as Per Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1 by Investigator Assessment for Combination A
Description: OR: complete response(CR) or partial response(PR)determined by investigator according to RECIST v1.1 from date of first dose of study treatment until date of first documentation of progressive disease(PD),confirmed by repeat assessments performed no less than 4 weeks after first response. CR: disappearance of target and non-target lesions, with exception of nodal disease and normalization of tumor markers. All nodes, target and non-target must have short axis measures less than (<)10 millimeter(mm). PR: >=30% decrease in sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of target lesions, taking as reference baseline sum of diameters. Non-target lesions must be non-PD. PD: >=20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to relative increase of 20%, sum must also demonstrate an absolute increase of at least 5mm, appearance of one or more new lesions was considered PD.
Time Frame: From start of the treatment until disease progression or death due to any cause, whichever occurred first (maximum up to 53 months approximately)
Population: The analysis population included all participants who received at least one dose of study drug. Participants were classified according to the study treatment actually received. If a participant received more than one treatment the participant was classified according to the first treatment received.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Combination A Phase 2 Melanoma: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCCHN: Utomilumab 100 mg + Avelumab | Combination A Phase 2 TNBC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 First Line (1L) NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 1L NSCLC: Utomilumab Then Utomilumab + Avelumab | Combination A Phase 2 1L NSCLC: Avelumab Then Utomilumab + Avelumab
Number analyzed (Participants) | 28 | 35 | 21 | 10 | 21 | 11 | 11
Percentage of participants | 10.7 [2.3 to 28.2] | 8.6 [1.8 to 23.1] | 14.3 [3.0 to 36.3] | 10.0 [0.3 to 44.5] | 4.8 [0.1 to 23.8] | 54.5 [23.4 to 83.3] | 18.2 [2.3 to 51.8]

7. Primary Outcome: Phase 2: Percentage of Participants With Confirmed OR as Per RECIST v 1.1 by Investigator Assessment for Combination B
Description: OR: CR or PR determined by investigator according to RECIST v1.1 from date of first dose of study treatment until date of first documentation of PD, confirmed by repeat assessments performed no less than 4 weeks after first response. CR: disappearance of target and non-target lesions, with exception of nodal disease and normalization of tumor markers. All nodes, target and non-target must have short axis measures <10 mm. PR: >=30% decrease in sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of target lesions, taking as reference baseline sum of diameters. Non-target lesions must be non-PD. PD: >=20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to relative increase of 20%, sum must also demonstrate an absolute increase of at least 5 mm, appearance of one or more new lesions was considered PD.
Time Frame: From start of the treatment until disease progression or death due to any cause, whichever occurred first (approximately 26 months)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Combination B Phase 2 NSCLC: PF-04518600 0.3 mg/kg + Avelumab | Combination B Phase 2 SCCHN: PF-04518600 0.3 mg/kg + Avelumab
Number analyzed (Participants) | 14 | 25
Percentage of participants | 14.3 [1.8 to 42.8] | 8.0 [1.0 to 26.0]

8. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Grade >= 3 TEAEs, Serious TEAEs and Treatment Related TEAEs: Combination A
Description: TEAEs are those events with onset dates occurring during the on-treatment period for the first time, or if the worsening of an event is during the on-treatment period. Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Per National Cancer Institute (NCI) CTCAE v4.03: Grade 3 (Severe) events=unacceptable or intolerable events, significantly interrupting usual daily activity, require systemic drug therapy/other treatment; Grade 4 (Life-threatening) events caused participant to be in imminent danger of death; Grade 5 (Death) events=death related to an AE. A serious AE (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in participant hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline up to 30 days after last dose of study treatment or the day before start day of new anti-cancer therapy (maximum of 6.5 years)
Population: The analysis population included all participants who received at least one dose of study drug. Participants were classified according to the study treatment actually received. If a participant received more than one study treatment, the participant were classified according to the first treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination A Phase 1b NSCLC: Utomilumab 500 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 20 mg + Avelumab | Combination A Phase 2 Melanoma: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCCHN: Utomilumab 100 mg + Avelumab | Combination A Phase 2 TNBC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 First Line (1L) NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 1L NSCLC: Utomilumab Then Utomilumab + Avelumab | Combination A Phase 2 1L NSCLC: Avelumab Then Utomilumab + Avelumab
Number analyzed (Participants) | 29 | 27 | 29 | 28 | 35 | 21 | 10 | 21 | 11 | 11
Participants
  TEAEs | 29 | 27 | 29 | 28 | 35 | 20 | 10 | 21 | 11 | 11
  Grade >=3 TEAEs | 15 | 13 | 18 | 13 | 19 | 9 | 7 | 12 | 8 | 6
  Serious TEAEs | 11 | 12 | 13 | 9 | 16 | 4 | 4 | 8 | 4 | 1
  Treatment related TEAEs | 22 | 22 | 25 | 23 | 26 | 15 | 8 | 19 | 10 | 9

9. Secondary Outcome: Number of Participants With TEAEs, Grade >= 3 TEAEs, Serious TEAEs and Treatment Related TEAEs: Combination B
Description: TEAEs are those events with onset dates occurring during the on-treatment period for the first time, or if the worsening of an event is during the on-treatment period. Treatment-related AEs was any untoward medical occurrence attributed to study drug in a participant who received study drug. Per NCI CTCAE v4.03: Grade 3 (Severe) events=unacceptable or intolerable events, significantly interrupting usual daily activity, require systemic drug therapy/other treatment; Grade 4 (Life-threatening) events caused participant to be in imminent danger of death; Grade 5 (Death) events=death related to an AE. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in participant hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline up to 30 days after last dose of study treatment or the day before start day of new anti-cancer therapy (maximum of 3.5 years)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Combination B Phase 1b: PF-04518600 0.3 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 1.0 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 3.0 mg/kg + Avelumab | Combination B Phase 2 NSCLC: PF-04518600 0.3 mg/kg + Avelumab | Combination B Phase 2 SCCHN: PF-04518600 0.3 mg/kg + Avelumab
Number analyzed (Participants) | 12 | 12 | 8 | 14 | 25
Participants
  TEAEs | 12 | 12 | 8 | 14 | 25
  Grade >=3 TEAEs | 4 | 6 | 4 | 7 | 13
  Serious TEAEs | 3 | 4 | 1 | 3 | 10
  Treatment related TEAEs | 7 | 7 | 7 | 12 | 14

10. Secondary Outcome: Number of Participants With TEAEs, Grade >= 3 TEAEs, Serious TEAEs and Treatment Related TEAEs: Combination C
Description: as for outcome 9
Time Frame: Baseline up to 30 days after last dose of study treatment or the day before start day of new anti-cancer therapy (maximum of 1.8 years)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Combination C Phase 1b: PD 0360324 50 mg + Avelumab | Combination C Phase 1b: PD 0360324 100 mg + Avelumab | Combination C Phase 1b: PD 0360324 150 mg + Avelumab
Number analyzed (Participants) | 10 | 8 | 6
Participants
  TEAEs | 9 | 8 | 6
  Grade >=3 TEAEs | 5 | 4 | 6
  Serious TEAEs | 4 | 3 | 4
  Treatment related TEAEs | 7 | 6 | 5

11. Secondary Outcome: Number of Participants With TEAEs, Grade >= 3 TEAEs, Serious TEAEs and Treatment Related TEAEs: Combination D
Description: as for outcome 9
Time Frame: Baseline up to 30 days after last dose of study treatment or the day before start day of new anti-cancer therapy (maximum of 4.3 years)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 1.0 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 1.0 mg/kg + Avelumab
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 11
Participants
  TEAEs | 12 | 12 | 12 | 12 | 12 | 11
  Grade >=3 TEAEs | 5 | 8 | 5 | 7 | 6 | 9
  Serious TEAEs | 2 | 3 | 4 | 5 | 4 | 5
  Treatment related TEAEs | 7 | 11 | 9 | 10 | 10 | 8

12. Secondary Outcome: Number of Participants With TEAEs, Grade >= 3 TEAEs, Serious TEAEs and Treatment Related TEAEs: Combination F
Description: as for outcome 9
Time Frame: Baseline up to 30 days after last dose of study treatment or the day before start day of new anti-cancer therapy (maximum of 3 years)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Combination F Phase 1b SCCHN: CMP-001 10 mg + Avelumab | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + Utomilumab 100 mg | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + PF-04518600 0.3 mg/kg
Number analyzed (Participants) | 6 | 7 | 7
Participants
  TEAEs | 6 | 7 | 7
  Grade >=3 TEAEs | 4 | 5 | 6
  Serious TEAEs | 2 | 4 | 4
  Treatment related TEAEs | 6 | 6 | 7

13. Secondary Outcome: Number of Participants With New Abnormal or Worsening Hematology Laboratory Test by Maximum Common Terminology Criteria for Adverse Events (CTCAE) Grade >=3: Combination A
Description: The laboratory results were graded according to the NCI CTCAE v4.03 severity grade. Grade 1=mild AE. Grade 2=moderate AE. Grade 3=severe AE. Grade 4=life-threatening consequences; urgent intervention indicated. Number of participants with new abnormal or worsening hematology laboratory test is presented." Participants with any grade >=3 is presented for following parameters: Anemia, lymphocyte count decreased, Platelet count decreased, neutrophil count decreased, and white blood cell decreased. Baseline is defined as the last assessment prior to the date/time of the first dose of study treatment.
Time Frame: Baseline up to end of treatment/withdrawal (maximum of 6.5 years)
Population: All participants who received at least one dose of study drug and who could be evaluated for CTCAE criteria for each parameter in each treatment group. Participants were classified according to study treatment actually received. If participant received more than one study treatment, participant was classified according to first treatment received. Here, "N''=number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination A Phase 1b NSCLC: Utomilumab 500 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 20 mg + Avelumab | Combination A Phase 2 Melanoma: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCCHN: Utomilumab 100 mg + Avelumab | Combination A Phase 2 TNBC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 First Line (1L) NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 1L NSCLC: Utomilumab Then Utomilumab + Avelumab | Combination A Phase 2 1L NSCLC: Avelumab Then Utomilumab + Avelumab
Number analyzed (Participants) | 28 | 27 | 29 | 28 | 34 | 21 | 10 | 21 | 11 | 11
Participants
  Participants with any grade >= 3 Anemia | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
  Participants with any grade >=3 Lymphocyte Count Decreased | 7 | 3 | 6 | 2 | 6 | 2 | 0 | 2 | 0 | 2
  Participants with any grade >= 3 Neutrophil Count Decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Participants with any grade >= 3 Platelet Count Decreased | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Participants with any grade >= 3 White Blood Cell Decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

14. Secondary Outcome: Number of Participants With New Abnormal or Worsening Hematology Laboratory Test by Maximum CTCAE Grade >=3: Combination B
Description: as for outcome 13
Time Frame: Baseline up to end of treatment/withdrawal (maximum of 3.5 years)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Combination B Phase 1b: PF-04518600 0.3 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 1.0 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 3.0 mg/kg + Avelumab | Combination B Phase 2 NSCLC: PF-04518600 0.3 mg/kg + Avelumab | Combination B Phase 2 SCCHN: PF-04518600 0.3 mg/kg + Avelumab
Number analyzed (Participants) | 12 | 12 | 8 | 14 | 24
Participants
  Participants with any grade >= 3 Anemia | 1 | 2 | 0 | 0 | 0
  Participants with any grade >=3 Lymphocyte Count Decreased | 1 | 3 | 1 | 3 | 8
  Participants with any grade >= 3 Neutrophil Count Decreased | 0 | 0 | 0 | 0 | 0
  Participants with any grade >= 3 Platelet Count Decreased | 0 | 0 | 0 | 1 | 0
  Participants with any grade >= 3 White Blood Cell Decreased | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With New Abnormal or Worsening Hematology Laboratory Test by Maximum CTCAE Grade >=3: Combination C
Description: as for outcome 13
Time Frame: Baseline up to end of treatment/withdrawal (maximum of 1.8 years)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Combination C Phase 1b: PD 0360324 50 mg + Avelumab | Combination C Phase 1b: PD 0360324 100 mg + Avelumab | Combination C Phase 1b: PD 0360324 150 mg + Avelumab
Number analyzed (Participants) | 10 | 8 | 6
Participants
  Participants with any grade >= 3 Anemia | 1 | 1 | 0
  Participants with any grade >=3 Lymphocyte Count Decreased | 1 | 1 | 1
  Participants with any grade >= 3 Neutrophil Count Decreased | 0 | 1 | 0
  Participants with any grade >= 3 Platelet Count Decreased | 0 | 0 | 0
  Participants with any grade >= 3 White Blood Cell Decreased | 0 | 1 | 0

16. Secondary Outcome: Number of Participants With New Abnormal or Worsening Hematology Laboratory Test by Maximum CTCAE Grade >=3: Combination D
Description: as for outcome 13
Time Frame: Baseline up to end of treatment/withdrawal (maximum of 4.3 years)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 1.0 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 1.0 mg/kg + Avelumab
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 12 | 11
Participants
  Participants with any grade >= 3 Anemia | 0 | 1 | 1 | 0 | 0 | 0
  Participants with any grade >=3 Lymphocyte Count Decreased | 3 | 6 | 6 | 2 | 3 | 1
  Participants with any grade >= 3 Neutrophil Count Decreased | 0 | 0 | 0 | 0 | 0 | 0
  Participants with any grade >= 3 Platelet Count Decreased | 0 | 0 | 1 | 0 | 1 | 0
  Participants with any grade >= 3 White Blood Cell Decreased | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With New Abnormal or Worsening Hematology Laboratory Test by Maximum CTCAE Grade >=3: Combination F
Description: as for outcome 13
Time Frame: Baseline up to end of treatment/withdrawal (maximum of 3 years)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Combination F Phase 1b SCCHN: CMP-001 10 mg + Avelumab | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + Utomilumab 100 mg | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + PF-04518600 0.3 mg/kg
Number analyzed (Participants) | 5 | 7 | 7
Participants
  Participants with any grade >= 3 Anemia | 0 | 2 | 2
  Participants with any grade >=3 Lymphocyte Count Decreased | 1 | 3 | 1
  Participants with any grade >= 3 Neutrophil Count Decreased | 1 | 0 | 0
  Participants with any grade >= 3 Platelet Count Decreased | 0 | 1 | 1
  Participants with any grade >= 3 White Blood Cell Decreased | 0 | 0 | 0

18. Secondary Outcome: Number of Participants With New Abnormal or Worsening Chemistry Laboratory Test Results During the On-Treatment Period by Maximum CTCAE Grade >=3: Combination A
Description: The laboratory results were graded according to the NCI CTCAE v4.03 severity grade. Grade 1=mild AE. Grade 2=moderate AE. Grade 3=severe AE. Grade 4=life-threatening consequences; urgent intervention indicated. Number of participants with new abnormal or worsening chemistry laboratory test is presented." Participants with any grade >=3 is presented for following parameters: Alanine aminotransferase increased, alkaline phosphatase increased, aspartate aminotransferase increased, blood bilirubin increased, creatinine increased, hyperglycemia, lipase increased and serum amylase increased. Baseline is defined as the last assessment prior to the date/time of the first dose of study treatment.
Time Frame: Baseline up to end of treatment/withdrawal (maximum of 6.5 years)
Population: All participants who received at least one dose of study drug and who could be evaluated for CTCAE criteria for each parameter in each treatment group. Participants were classified according to study treatment actually received. If participant received more than one study treatment, participant was classified according to first treatment received. Here, "N''=number of participants evaluable for this outcome measure, where n=number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination A Phase 1b NSCLC: Utomilumab 500 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 20 mg + Avelumab | Combination A Phase 2 Melanoma: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCCHN: Utomilumab 100 mg + Avelumab | Combination A Phase 2 TNBC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 First Line (1L) NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 1L NSCLC: Utomilumab Then Utomilumab + Avelumab | Combination A Phase 2 1L NSCLC: Avelumab Then Utomilumab + Avelumab
Number analyzed (Participants) | 28 | 27 | 29 | 28 | 34 | 21 | 10 | 21 | 11 | 11
Participants
  Participants with any grade >= 3 Alanine Aminotransferase Increased | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Participants with any grade >= 3 Alkaline Phosphatase Increased | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Participants with any grade >= 3 Aspartate Aminotransferase Increased | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
  Participants with any grade >= 3 Blood Bilirubin Increased | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Participants with any grade >= 3 Creatinine Increased | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Participants with any grade >= 3 Hyperglycemia | 2 | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 1 | 3
  Participants with any grade >= 3 Lipase Increased: number analyzed (Participants) | 28 | 27 | 29 | 28 | 34 | 21 | 9 | 20 | 11 | 11
  Participants with any grade >= 3 Lipase Increased | 2 | 0 | 2 | 4 | 1 | 2 | 0 | 1 | 0 | 2
  Participants with any grade >= 3 Serum Amylase Increased: number analyzed (Participants) | 28 | 27 | 29 | 28 | 34 | 21 | 9 | 20 | 11 | 11
  Participants with any grade >= 3 Serum Amylase Increased | 2 | 1 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 1

19. Secondary Outcome: Number of Participants With New Abnormal or Worsening Chemistry Laboratory Test Results During the On-Treatment Period by Maximum CTCAE Grade >=3: Combination B
Description: as for outcome 18
Time Frame: Baseline up to end of treatment/withdrawal (maximum of 3.5 years)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Combination B Phase 1b: PF-04518600 0.3 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 1.0 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 3.0 mg/kg + Avelumab | Combination B Phase 2 NSCLC: PF-04518600 0.3 mg/kg + Avelumab | Combination B Phase 2 SCCHN: PF-04518600 0.3 mg/kg + Avelumab
Number analyzed (Participants) | 12 | 12 | 8 | 14 | 24
Participants
  Participants with any grade >= 3 Alanine Aminotransferase Increased | 0 | 0 | 0 | 0 | 0
  Participants with any grade >= 3 Alkaline Phosphatase Increased | 1 | 0 | 0 | 0 | 0
  Participants with any grade >= 3 Aspartate Aminotransferase Increased | 1 | 0 | 0 | 0 | 0
  Participants with any grade >= 3 Blood Bilirubin Increased | 0 | 0 | 0 | 0 | 0
  Participants with any grade >= 3 Creatinine Increased | 0 | 0 | 0 | 0 | 1
  Participants with any grade >= 3 Hyperglycemia | 1 | 0 | 0 | 0 | 2
  Participants with any grade >= 3 Lipase Increased | 1 | 1 | 1 | 4 | 5
  Participants with any grade >= 3 Serum Amylase Increased | 0 | 0 | 0 | 1 | 0

20. Secondary Outcome: Number of Participants With New Abnormal or Worsening Chemistry Laboratory Test Results During the On-Treatment Period by Maximum CTCAE Grade >=3: Combination C
Description: as for outcome 18
Time Frame: Baseline up to end of treatment/withdrawal (maximum of 1.8 years)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Combination C Phase 1b: PD 0360324 50 mg + Avelumab | Combination C Phase 1b: PD 0360324 100 mg + Avelumab | Combination C Phase 1b: PD 0360324 150 mg + Avelumab
Number analyzed (Participants) | 10 | 8 | 6
Participants
  Participants with any grade >= 3 Alanine Aminotransferase Increased | 0 | 0 | 2
  Participants with any grade >= 3 Alkaline Phosphatase Increased | 0 | 0 | 0
  Participants with any grade >= 3 Aspartate Aminotransferase Increased | 0 | 0 | 1
  Participants with any grade >= 3 Blood Bilirubin Increased | 0 | 0 | 0
  Participants with any grade >= 3 Creatinine Increased | 0 | 0 | 0
  Participants with any grade >= 3 Hyperglycemia | 2 | 0 | 2
  Participants with any grade >= 3 Lipase Increased | 1 | 3 | 2
  Participants with any grade >= 3 Serum Amylase Increased | 0 | 1 | 0

21. Secondary Outcome: Number of Participants With New Abnormal or Worsening Chemistry Laboratory Test Results During the On-Treatment Period by Maximum CTCAE Grade >=3: Combination D
Description: as for outcome 18
Time Frame: Baseline up to end of treatment/withdrawal (maximum of 4.3 years)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 1.0 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 1.0 mg/kg + Avelumab
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 12 | 11
Participants
  Participants with any grade >= 3 Alanine Aminotransferase Increased | 0 | 0 | 0 | 1 | 0 | 1
  Participants with any grade >= 3 Alkaline Phosphatase Increased | 0 | 0 | 0 | 0 | 0 | 1
  Participants with any grade >= 3 Aspartate Aminotransferase Increased | 0 | 0 | 0 | 1 | 0 | 1
  Participants with any grade >= 3 Blood Bilirubin Increased | 0 | 0 | 0 | 0 | 0 | 1
  Participants with any grade >= 3 Creatinine Increased | 0 | 0 | 0 | 0 | 0 | 0
  Participants with any grade >= 3 Hyperglycemia | 1 | 1 | 0 | 1 | 2 | 1
  Participants with any grade >= 3 Lipase Increased | 0 | 3 | 2 | 2 | 2 | 1
  Participants with any grade >= 3 Serum Amylase Increased | 0 | 0 | 0 | 0 | 0 | 1

22. Secondary Outcome: Number of Participants With New Abnormal or Worsening Chemistry Laboratory Test Results During the On-Treatment Period by Maximum CTCAE Grade >=3: Combination F
Description: as for outcome 18
Time Frame: Baseline up to end of treatment/withdrawal (maximum of 3 years)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Combination F Phase 1b SCCHN: CMP-001 10 mg + Avelumab | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + Utomilumab 100 mg | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + PF-04518600 0.3 mg/kg
Number analyzed (Participants) | 5 | 7 | 7
Participants
  Participants with any grade >= 3 Alanine Aminotransferase Increased | 0 | 0 | 0
  Participants with any grade >= 3 Alkaline Phosphatase Increased | 0 | 0 | 0
  Participants with any grade >= 3 Aspartate Aminotransferase Increased | 0 | 1 | 0
  Participants with any grade >= 3 Blood Bilirubin Increased | 0 | 0 | 0
  Participants with any grade >= 3 Creatinine Increased | 0 | 0 | 0
  Participants with any grade >= 3 Hyperglycemia | 0 | 0 | 1
  Participants with any grade >= 3 Lipase Increased | 1 | 0 | 1
  Participants with any grade >= 3 Serum Amylase Increased | 1 | 0 | 0

23. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Avelumab in Combination A
Description: Cmax is maximum observed plasma concentration.
Time Frame: 1-hour post-dose (at end of infusion) on Day 1,15 of Cycle 1; Day 8 of Cycle 1 (non-dosing); Day 1 of Cycle 2, 4, 6, 10. For ''Phase 2 1L NSCLC: Utomilumab then Utomilumab + Avelumab'' reporting group: Day 1 of Cycle 2, 4, 6, 10
Population: All participants who received at least one dose of study drug and who had at least one of the PK concentrations for Avelumab, Utomilumab, PD 0360324, PF-04518600. Here, "Number of participants analyzed'' signifies number of participants evaluable for this outcome measure, where "Number Analyzed" signifies number of participants evaluable for specified time points. For ''Phase 2 1L NSCLC: Utomilumab then Utomilumab + Avelumab'' reporting group PK sampling started from Cycle 2 Day 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Combination A Phase 1b NSCLC: Utomilumab 500 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 20 mg + Avelumab | Combination A Phase 2 Melanoma: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCCHN: Utomilumab 100 mg + Avelumab | Combination A Phase 2 TNBC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 First Line (1L) NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 1L NSCLC: Utomilumab Then Utomilumab + Avelumab | Combination A Phase 2 1L NSCLC: Avelumab Then Utomilumab + Avelumab
Number analyzed (Participants) | 28 | 27 | 29 | 26 | 29 | 21 | 9 | 20 | 7 | 10
Nanogram per milliliter
  Cycle 1/Day1-1 Hour/End Of Infusion (EOI): number analyzed (Participants) | 22 | 27 | 24 | 24 | 29 | 19 | 9 | 16 | 0 | 9
  Cycle 1/Day1-1 Hour/End Of Infusion (EOI) | 232.6 (39) | 219.0 (26) | 231.2 (37) | 262.0 (56) | 209.0 (31) | 215.5 (26) | 284.2 (16) | 218.6 (29) |  | 194.4 (27)
  Cycle 1/Day8-168 Hour: number analyzed (Participants) | 28 | 26 | 29 | 26 | 27 | 21 | 8 | 20 | 0 | 10
  Cycle 1/Day8-168 Hour | 63.60 (52) | 59.86 (65) | 61.49 (84) | 73.57 (78) | 69.14 (43) | 60.03 (33) | 51.85 (36) | 45.69 (25) |  | 34.46 (45)
  Cycle 1/Day15-1 Hour/EOI: number analyzed (Participants) | 18 | 21 | 24 | 24 | 26 | 15 | 5 | 12 | 0 | 9
  Cycle 1/Day15-1 Hour/EOI | 212.1 (84) | 226.1 (26) | 253.6 (31) | 279.4 (33) | 238.9 (26) | 241.9 (29) | 324.6 (27) | 221.2 (23) |  | 193.7 (24)
  Cycle 2/Day1-1 Hour/EOI: number analyzed (Participants) | 16 | 20 | 20 | 22 | 28 | 11 | 4 | 12 | 7 | 6
  Cycle 2/Day1-1 Hour/EOI | 276.0 (33) | 229.0 (33) | 267.9 (31) | 255.5 (72) | 223.4 (30) | 292.0 (18) | 302.5 (23) | 222.0 (29) | 200.1 (20) | 203.3 (16)
  Cycle 4/Day1-1 Hour/EOI: number analyzed (Participants) | 8 | 8 | 10 | 10 | 15 | 6 | 1 | 6 | 5 | 6
  Cycle 4/Day1-1 Hour/EOI | 258.4 (18) | 232.8 (20) | 285.6 (16) | 303.1 (79) | 209.5 (22) | 283.0 (27) | 215.0 (NA) — Geometric Coefficient of Variation was not estimable as there was only 1 participant analyzed. | 273.5 (18) | 206.9 (13) | 97.46 (237)
  Cycle 6/Day1-1 Hour/EOI: number analyzed (Participants) | 8 | 6 | 5 | 5 | 13 | 5 | 2 | 4 | 5 | 4
  Cycle 6/Day1-1 Hour/EOI | 248.4 (32) | 211.1 (20) | 193.2 (121) | 512.8 (126) | 217.1 (28) | 305.9 (18) | 332.9 (3) | 275.2 (42) | 208.3 (17) | 218.3 (11)
  Cycle 10/Day1-1 Hour/EOI: number analyzed (Participants) | 5 | 4 | 4 | 4 | 5 | 2 | 1 | 1 | 3 | 3
  Cycle 10/Day1-1 Hour/EOI | 230.0 (48) | 180.5 (39) | 328.1 (14) | 248.4 (14) | 228.1 (20) | 187.2 (73) | 335.0 (NA) — Geometric Coefficient of Variation was not estimable as there was only 1 participant analyzed. | 102.0 (NA) — Geometric Coefficient of Variation was not estimable as there was only 1 participant analyzed. | 251.2 (14) | 89.72 (374)

24. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Utomilumab in Combination A
Description: Cmax is maximum observed plasma concentration.
Time Frame: 1-hour post-infusion (at end of infusion) on Day 1 of Cycle 1,3,5,8,12; Day 8 of Cycle 1 (non-dosing). For ''Phase 2 1L NSCLC: Avelumab then Utomilumab + Avelumab'' reporting group: Day 1 of Cycle 3,5,8,12
Population: All participants who received at least one dose of study drug and who had at least one of the PK concentrations for Avelumab, Utomilumab, PD 0360324, PF-04518600. Here, "Number of participants analyzed'' signifies number of participants evaluable for this outcome measure, where "Number Analyzed" signifies number of participants evaluable for specified time points. For participants of ''Phase 2 1L NSCLC: Avelumab then Utomilumab + Avelumab'' reporting group PK sampling started from Cycle 3 Day 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Combination A Phase 1b NSCLC: Utomilumab 500 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 20 mg + Avelumab | Combination A Phase 2 Melanoma: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCCHN: Utomilumab 100 mg + Avelumab | Combination A Phase 2 TNBC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 First Line (1L) NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 1L NSCLC: Utomilumab Then Utomilumab + Avelumab | Combination A Phase 2 1L NSCLC: Avelumab Then Utomilumab + Avelumab
Number analyzed (Participants) | 28 | 27 | 29 | 28 | 32 | 21 | 10 | 20 | 10 | 7
Nanogram per milliliter
  Cycle 1/Day1-1 Hour/EOI: number analyzed (Participants) | 27 | 27 | 28 | 28 | 32 | 21 | 10 | 19 | 9 | 0
  Cycle 1/Day1-1 Hour/EOI | 106500 (31) | 27250 (30) | 4673 (45) | 23520 (34) | 26960 (24) | 23780 (39) | 20790 (39) | 20570 (28) | 26020 (35) |
  Cycle 1/Day8-168 Hour: number analyzed (Participants) | 28 | 26 | 29 | 26 | 27 | 21 | 8 | 20 | 10 | 0
  Cycle 1/Day8-168 Hour | 15940 (126) | 4584 (93) | 1070 (38) | 5740 (73) | 7344 (60) | 8692 (56) | 5036 (35) | 6671 (41) | 7185 (135) |
  Cycle 3/Day1-1 Hour/EOI: number analyzed (Participants) | 16 | 12 | 21 | 14 | 16 | 8 | 3 | 9 | 8 | 7
  Cycle 3/Day1-1 Hour/EOI | 132000 (19) | 26250 (19) | 6446 (58) | 26210 (26) | 28880 (31) | 35950 (21) | 15170 (26) | 20190 (66) | 27710 (35) | 26710 (21)
  Cycle 5/Day1-1 Hour/EOI: number analyzed (Participants) | 10 | 6 | 7 | 8 | 14 | 7 | 3 | 5 | 6 | 7
  Cycle 5/Day1-1 Hour/EOI | 134800 (29) | 26470 (70) | 5800 (48) | 32630 (51) | 28370 (25) | 28000 (36) | 11270 (98) | 19440 (48) | 25650 (30) | 15410 (141)
  Cycle 8/Day1-1 Hour/EOI: number analyzed (Participants) | 7 | 4 | 4 | 6 | 5 | 4 | 2 | 2 | 6 | 5
  Cycle 8/Day1-1 Hour/EOI | 121800 (28) | 13340 (951) | 6067 (20) | 38930 (85) | 19870 (92) | 20710 (38) | 20710 (22) | 16750 (34) | 21680 (22) | 18080 (89)
  Cycle 12/Day1-1 Hour/EOI: number analyzed (Participants) | 6 | 3 | 4 | 5 | 2 | 3 | 0 | 1 | 3 | 3
  Cycle 12/Day1-1 Hour/EOI | 124800 (30) | 19800 (62) | 6892 (26) | 44690 (225) | 20460 (8) | 27030 (28) |  | 12900 (NA) — Geometric Coefficient of Variation was not estimable as there was only 1 participant analyzed. | 20730 (33) | 24060 (1)

25. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Avelumab and PF-04518600 in Combination B
Description: Cmax is maximum observed plasma concentration.
Time Frame: 1-hour post-dose on Day 1,15 of Cycle 1; Day 8 of Cycle 1 (non-dosing); Day 1 of Cycle 2, 4, 6 and Cycle 10
Population: Pharmacokinetic (PK) analysis set included all participants who had received at least one dose of study drug and who had at least one of the PK concentrations of interest for Avelumab, Utomilumab, PD 0360324, PF-04518600. Here, "Number of participants analyzed'' signifies number of participants evaluable for this outcome measure, where "Number Analyzed" signifies number of participants evaluable for specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Combination B Phase 1b: PF-04518600 0.3 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 1.0 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 3.0 mg/kg + Avelumab | Combination B Phase 2 NSCLC: PF-04518600 0.3 mg/kg + Avelumab | Combination B Phase 2 SCCHN: PF-04518600 0.3 mg/kg + Avelumab
Number analyzed (Participants) | 12 | 12 | 8 | 13 | 23
Nanogram per milliliter
  Avelumab Cycle 1/Day1-1 Hour/EOI: number analyzed (Participants) | 9 | 12 | 7 | 11 | 22
  Avelumab Cycle 1/Day1-1 Hour/EOI | 220.6 (26) | 257.6 (65) | 213.7 (30) | 219.8 (22) | 178.4 (31)
  Avelumab Cycle 1/Day8-168 Hour: number analyzed (Participants) | 11 | 11 | 8 | 13 | 23
  Avelumab Cycle 1/Day8-168 Hour | 54.00 (51) | 42.66 (50) | 49.85 (45) | 50.86 (35) | 47.68 (33)
  Avelumab Cycle 1/Day15-1 Hour/EOI: number analyzed (Participants) | 7 | 10 | 6 | 9 | 20
  Avelumab Cycle 1/Day15-1 Hour/EOI | 241.9 (23) | 240.3 (17) | 228.7 (33) | 235.5 (29) | 180.3 (68)
  Avelumab Cycle 2/Day1-1 Hour/EOI: number analyzed (Participants) | 8 | 8 | 6 | 10 | 20
  Avelumab Cycle 2/Day1-1 Hour/EOI | 242.8 (22) | 256.2 (18) | 277.1 (27) | 249.1 (22) | 188.4 (22)
  Avelumab Cycle 4/Day1-1 Hour/EOI: number analyzed (Participants) | 3 | 2 | 2 | 6 | 11
  Avelumab Cycle 4/Day1-1 Hour/EOI | 223.9 (19) | 204.1 (44) | 254.4 (10) | 184.9 (31) | 205.6 (21)
  Avelumab Cycle 6/Day1-1 Hour/EOI: number analyzed (Participants) | 0 | 1 | 0 | 3 | 5
  Avelumab Cycle 6/Day1-1 Hour/EOI |  | 143.0 (NA) — Geometric Coefficient of Variation was not estimable as there was only 1 participant analyzed. |  | 280.6 (18) | 137.0 (110)
  Avelumab Cycle 10/Day1-1 Hour/EOI: number analyzed (Participants) | 0 | 0 | 0 | 1 | 4
  Avelumab Cycle 10/Day1-1 Hour/EOI |  |  |  | 231.0 (NA) — Geometric Coefficient of Variation was not estimable as there was only 1 participant analyzed. | 197.2 (13)
  PF- 04518600 Cycle 1/Day1-1 Hour/EOI: number analyzed (Participants) | 12 | 12 | 7 | 12 | 23
  PF- 04518600 Cycle 1/Day1-1 Hour/EOI | 6413 (21) | 21560 (25) | 74090 (13) | 6919 (28) | 6085 (37)
  PF-04518600 Cycle 1/Day8-168 Hour: number analyzed (Participants) | 11 | 11 | 8 | 13 | 23
  PF-04518600 Cycle 1/Day8-168 Hour | 2669 (51) | 9427 (25) | 31650 (34) | 3131 (32) | 2631 (28)
  PF-04518600 Cycle 1/Day15-1 Hour/EOI: number analyzed (Participants) | 9 | 10 | 7 | 13 | 19
  PF-04518600 Cycle 1/Day15-1 Hour/EOI | 5969 (77) | 27460 (24) | 96640 (22) | 6697 (71) | 7173 (35)
  PF-04518600 Cycle 2/Day1-1 Hour/EOI: number analyzed (Participants) | 11 | 8 | 7 | 12 | 23
  PF-04518600 Cycle 2/Day1-1 Hour/EOI | 7776 (33) | 31880 (16) | 104100 (56) | 9212 (30) | 7627 (25)
  PF-04518600 Cycle 4/Day1-1 Hour/EOI: number analyzed (Participants) | 3 | 0 | 3 | 9 | 12
  PF-04518600 Cycle 4/Day1-1 Hour/EOI | 8792 (43) |  | 155000 (20) | 11730 (61) | 10180 (36)
  PF-04518600 Cycle 6/Day1-1 Hour/EOI: number analyzed (Participants) | 0 | 1 | 0 | 6 | 5
  PF-04518600 Cycle 6/Day1-1 Hour/EOI |  | 32000 (NA) — Geometric Coefficient of Variation was not estimable as there was only 1 participant analyzed. |  | 14020 (27) | 9753 (10)
  PF-04518600 Cycle 10/Day1-1 Hour/EOI: number analyzed (Participants) | 0 | 0 | 0 | 2 | 4
  PF-04518600 Cycle 10/Day1-1 Hour/EOI |  |  |  | 14060 (16) | 10660 (18)

26. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Avelumab and PD 0360324 in Combination C
Description: Cmax is maximum observed plasma concentration.
Time Frame: 1 hour (i.e. at the end of infusion) post-dose on Day 1,15 of Cycle 1; Day 8 of Cycle 1 (non-dosing); Day 1 of Cycle 2, 4, 6 and Cycle 10
Population: PK analysis set included all participants who had received at least one dose of study drug and who had at least one of the PK concentrations of interest for Avelumab, Utomilumab, PD 0360324, PF-04518600. Here, "Number of participants analyzed'' signifies number of participants evaluable for this outcome measure, where "Number Analyzed" signifies number of participants evaluable for specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Combination C Phase 1b: PD 0360324 50 mg + Avelumab | Combination C Phase 1b: PD 0360324 100 mg + Avelumab | Combination C Phase 1b: PD 0360324 150 mg + Avelumab
Number analyzed (Participants) | 10 | 7 | 6
Nanogram per milliliter
  Avelumab Cycle 1/Day1-1 Hour/EOI: number analyzed (Participants) | 9 | 7 | 2
  Avelumab Cycle 1/Day1-1 Hour/EOI | 217.0 (13) | 209.9 (34) | 247.9 (18)
  Avelumab Cycle 1/Day8-168 Hour: number analyzed (Participants) | 9 | 7 | 6
  Avelumab Cycle 1/Day8-168 Hour | 53.39 (31) | 63.12 (25) | 47.89 (28)
  Avelumab Cycle 1/Day15-1 Hour/EOI: number analyzed (Participants) | 8 | 7 | 3
  Avelumab Cycle 1/Day15-1 Hour/EOI | 233.8 (26) | 277.4 (20) | 263.6 (33)
  Avelumab Cycle 2/Day1-1 Hour/EOI: number analyzed (Participants) | 6 | 5 | 3
  Avelumab Cycle 2/Day1-1 Hour/EOI | 253.7 (15) | 295.2 (30) | 254.0 (20)
  Avelumab Cycle 4/Day1-1 Hour/EOI: number analyzed (Participants) | 2 | 2 | 2
  Avelumab Cycle 4/Day1-1 Hour/EOI | 242.0 (24) | 331.1 (29) | 304.8 (44)
  Avelumab Cycle 6/Day1-1 Hour/EOI: number analyzed (Participants) | 2 | 2 | 1
  Avelumab Cycle 6/Day1-1 Hour/EOI | 248.2 (17) | 292.4 (17) | 270.0 (NA) — Geometric Coefficient of Variation was not estimable as there was only 1 participant analyzed.
  Avelumab Cycle 10/Day1-1 Hour/EOI: number analyzed (Participants) | 0 | 1 | 0
  Avelumab Cycle 10/Day1-1 Hour/EOI |  | 318.0 (NA) — Geometric Coefficient of Variation was not estimable as there was only 1 participant analyzed. |
  PD 0360324 Cycle 1/Day1-30 Minutes (Min)/EOI: number analyzed (Participants) | 10 | 5 | 5
  PD 0360324 Cycle 1/Day1-30 Minutes (Min)/EOI | 17570 (22) | 34420 (55) | 38200 (44)
  PD 0360324 Cycle 1/Day8-168 Hour: number analyzed (Participants) | 9 | 6 | 6
  PD 0360324 Cycle 1/Day8-168 Hour | 1324 (109) | 8846 (43) | 6598 (47)
  PD 0360324 Cycle 1/Day15-30 min/EOI: number analyzed (Participants) | 9 | 6 | 5
  PD 0360324 Cycle 1/Day15-30 min/EOI | 16620 (27) | 32550 (29) | 46130 (51)
  PD 0360324 Cycle 2/Day1-30 min/EOI: number analyzed (Participants) | 8 | 6 | 5
  PD 0360324 Cycle 2/Day1-30 min/EOI | 17050 (20) | 11690 (1072) | 57420 (16)
  PD 0360324 Cycle 4/Day1-30 min/EOI: number analyzed (Participants) | 2 | 2 | 5
  PD 0360324 Cycle 4/Day1-30 min/EOI | 17700 (2) | 27060 (8) | 43650 (51)
  PD 0360324 Cycle 6/Day1-30 min/EOI: number analyzed (Participants) | 2 | 2 | 3
  PD 0360324 Cycle 6/Day1-30 min/EOI | 15590 (12) | 35140 (8) | 58620 (27)
  PD 0360324 Cycle 10/Day1-30 min/EOI: number analyzed (Participants) | 0 | 1 | 2
  PD 0360324 Cycle 10/Day1-30 min/EOI |  | 33100 (NA) — Geometric Coefficient of Variation was not estimable as there was only 1 participant analyzed. | 3216 (11668)

27. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Avelumab in Combination D
Description: Cmax is maximum observed plasma concentration.
Time Frame: 1 hour post-dose (at end of infusion) on Days 1 and 15 of Cycle 1; Day 8 of Cycle 1 (non-dosing); Pre-dose and 1 hour post-dose on Day 1 of Cycle 2, 4, 6, 10
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 1.0 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 1.0 mg/kg + Avelumab
Number analyzed (Participants) | 11 | 12 | 12 | 9 | 12 | 10
Nanogram per milliliter
  Cycle 1/Day1-1 Hour/EOI: number analyzed (Participants) | 10 | 11 | 12 | 8 | 12 | 10
  Cycle 1/Day1-1 Hour/EOI | 158.3 (26) | 188.2 (26) | 200.8 (22) | 185.1 (38) | 187.4 (18) | 174.2 (32)
  Cycle 1/Day8-168 Hour: number analyzed (Participants) | 11 | 12 | 12 | 9 | 12 | 9
  Cycle 1/Day8-168 Hour | 46.74 (46) | 37.71 (20) | 39.14 (24) | 41.96 (24) | 41.32 (24) | 36.07 (36)
  Cycle 1/Day15-1 Hour/EOI: number analyzed (Participants) | 11 | 9 | 12 | 5 | 11 | 7
  Cycle 1/Day15-1 Hour/EOI | 201.8 (20) | 124.1 (136) | 150.8 (91) | 167.3 (17) | 217.2 (20) | 80.14 (1114)
  Cycle 2/Day1-1 Hour/EOI: number analyzed (Participants) | 11 | 7 | 11 | 5 | 9 | 7
  Cycle 2/Day1-1 Hour/EOI | 200.4 (18) | 190.9 (23) | 149.2 (143) | 142.9 (42) | 228.5 (18) | 175.1 (24)
  Cycle 4/Day1-1 Hour/EOI: number analyzed (Participants) | 3 | 4 | 6 | 3 | 5 | 3
  Cycle 4/Day1-1 Hour/EOI | 188.9 (30) | 210.0 (23) | 193.9 (29) | 192.8 (6) | 223.2 (16) | 178.7 (25)
  Cycle 6/Day1-1 Hour/EOI: number analyzed (Participants) | 4 | 4 | 4 | 2 | 2 | 3
  Cycle 6/Day1-1 Hour/EOI | 216.7 (25) | 198.8 (34) | 208.2 (13) | 161.0 (4) | 217.1 (8) | 193.3 (19)
  Cycle 10/Day1-1 Hour/EOI: number analyzed (Participants) | 3 | 3 | 3 | 2 | 1 | 2
  Cycle 10/Day1-1 Hour/EOI | 203.7 (10) | 196.0 (53) | 194.5 (26) | 182.0 (2) | 268.0 (NA) — Geometric Coefficient of Variation was not estimable as there was only 1 participant analyzed. | 229.1 (34)

28. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Utomilumab in Combination D
Description: Cmax is maximum observed plasma concentration.
Time Frame: 1 hour (at end of infusion) post-dose on Day 1 of Cycles 1, 3, 5, 8 and Cycle 12; Days 8 of Cycle 1 (non-dosing)
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 1.0 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 1.0 mg/kg + Avelumab
Number analyzed (Participants) | 12 | 12 | 12 | 11 | 12 | 11
Nanogram per milliliter
  Cycle 1/Day1-1 Hour/EOI: number analyzed (Participants) | 12 | 10 | 12 | 11 | 12 | 11
  Cycle 1/Day1-1 Hour/EOI | 3370 (39) | 8935 (67) | 3751 (78) | 4919 (104) | 2155 (79) | 9567 (22)
  Cycle 1/Day8-168 Hour: number analyzed (Participants) | 11 | 12 | 12 | 9 | 12 | 9
  Cycle 1/Day8-168 Hour | 1406 (44) | 3066 (22) | 1043 (45) | 2437 (85) | 1318 (34) | 2940 (78)
  Cycle 3/Day1-1 Hour/EOI: number analyzed (Participants) | 5 | 5 | 8 | 6 | 7 | 5
  Cycle 3/Day1-1 Hour/EOI | 2413 (14) | 11820 (47) | 3953 (51) | 9471 (46) | 2669 (116) | 8877 (12)
  Cycle 5/Day1-1 Hour/EOI: number analyzed (Participants) | 4 | 5 | 5 | 1 | 4 | 4
  Cycle 5/Day1-1 Hour/EOI | 3477 (51) | 14310 (19) | 2694 (123) | 7500 (NA) — Geometric Coefficient of Variation was not estimable as there was only 1 participant analyzed. | 2475 (56) | 8029 (21)
  Cycle 8/Day1-1 Hour/EOI: number analyzed (Participants) | 2 | 4 | 4 | 2 | 2 | 2
  Cycle 8/Day1-1 Hour/EOI | 2596 (8) | 3354 (374) | 3202 (126) | 14790 (24) | 2028 (33) | 5542 (71)
  Cycle 12/Day1-1 Hour/EOI: number analyzed (Participants) | 2 | 4 | 2 | 2 | 1 | 0
  Cycle 12/Day1-1 Hour/EOI | 2460 (1) | 13400 (9) | 3422 (51) | 13220 (39) | 1120 (NA) — Geometric Coefficient of Variation was not estimable as there was only 1 participant analyzed. |

29. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-04518600 in Combination D
Description: Cmax is maximum observed plasma concentration.
Time Frame: 1 hour post-infusion (at end of infusion) on Day 1 and 15 of Cycle 1; Day 8 of Cycle 1 (non-dosing); Day 1 of Cycle 2, 4, 6 and Cycle 10
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 1.0 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 1.0 mg/kg + Avelumab
Number analyzed (Participants) | 11 | 12 | 12 | 12 | 12 | 11
Nanogram per milliliter
  Cycle 1/Day1-1 Hour/End Of Infusion (EOI): number analyzed (Participants) | 10 | 12 | 11 | 12 | 12 | 11
  Cycle 1/Day1-1 Hour/End Of Infusion (EOI) | 1698 (51) | 1714 (24) | 5224 (58) | 4417 (59) | 18250 (30) | 17770 (33)
  Cycle 1/Day8-168 Hour: number analyzed (Participants) | 11 | 12 | 12 | 9 | 12 | 8
  Cycle 1/Day8-168 Hour | 695.1 (26) | 589.5 (41) | 2379 (30) | 2139 (31) | 9717 (15) | 7700 (35)
  Cycle 1/Day15-1 Hour/EOI: number analyzed (Participants) | 11 | 11 | 12 | 8 | 12 | 7
  Cycle 1/Day15-1 Hour/EOI | 1841 (65) | 1823 (35) | 6595 (26) | 8559 (68) | 24470 (23) | 23330 (22)
  Cycle 2/Day1-1 Hour/EOI: number analyzed (Participants) | 8 | 8 | 11 | 7 | 8 | 7
  Cycle 2/Day1-1 Hour/EOI | 2278 (24) | 1901 (22) | 7497 (39) | 7373 (18) | 25890 (50) | 25180 (29)
  Cycle 4/Day1-1 Hour/EOI: number analyzed (Participants) | 5 | 5 | 5 | 3 | 7 | 3
  Cycle 4/Day1-1 Hour/EOI | 2711 (44) | 2453 (34) | 9984 (39) | 7279 (29) | 36930 (14) | 39590 (26)
  Cycle 6/Day1-1 Hour/EOI: number analyzed (Participants) | 4 | 5 | 3 | 2 | 4 | 3
  Cycle 6/Day1-1 Hour/EOI | 2633 (27) | 2704 (26) | 13340 (27) | 6637 (20) | 34540 (24) | 36190 (20)
  Cycle 10/Day1-1 Hour/EOI: number analyzed (Participants) | 3 | 4 | 4 | 2 | 2 | 2
  Cycle 10/Day1-1 Hour/EOI | 2741 (20) | 2685 (50) | 11130 (44) | 9026 (61) | 44170 (16) | 39190 (43)

30. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Avelumab in Combination F
Description: Cmax is maximum observed plasma concentration.
Time Frame: 1-hour post-infusion (i.e. at the end of infusion) on Days 1 and 15 of Cycle 1 (non-dosing); Day 1 of Cycles 2, 4, 6 and Cycle 10
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Combination F Phase 1b SCCHN: CMP-001 10 mg + Avelumab | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + Utomilumab 100 mg | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + PF-04518600 0.3 mg/kg
Number analyzed (Participants) | 6 | 6 | 6
Nanogram per milliliter
  Cycle 1/Day1-1 Hour/EOI: number analyzed (Participants) | 6 | 5 | 6
  Cycle 1/Day1-1 Hour/EOI | 161.2 (14) | 166.1 (15) | 180.7 (49)
  Cycle 1/Day15-1 Hour/EOI: number analyzed (Participants) | 5 | 6 | 5
  Cycle 1/Day15-1 Hour/EOI | 182.6 (11) | 171.2 (27) | 151.6 (16)
  Cycle 2/Day1-1 Hour/EOI: number analyzed (Participants) | 5 | 5 | 4
  Cycle 2/Day1-1 Hour/EOI | 165.5 (10) | 176.7 (22) | 171.0 (26)
  Cycle 4/Day1-1 Hour/EOI: number analyzed (Participants) | 2 | 3 | 0
  Cycle 4/Day1-1 Hour/EOI | 185.0 (24) | 203.9 (27) |
  Cycle 6/Day1-1 Hour/EOI: number analyzed (Participants) | 1 | 1 | 0
  Cycle 6/Day1-1 Hour/EOI | 229.0 (NA) — Geometric Coefficient of Variation was not estimable as there was only 1 participant analyzed. | 174.0 (NA) — Geometric Coefficient of Variation was not estimable as there was only 1 participant analyzed. |
  Cycle 10/Day1-1 Hour/EOI: number analyzed (Participants) | 1 | 0 | 0
  Cycle 10/Day1-1 Hour/EOI | 191.0 (NA) — Geometric Coefficient of Variation was not estimable as there was only 1 participant analyzed. |  |

31. Secondary Outcome: Pre-Dose Observed Plasma Concentration (Ctrough) of Avelumab in Combination A
Description: Ctrough is steady-state pre-dose concentration.
Time Frame: Pre-dose on Days 1 and 15 of Cycle 1, Day 8 of Cycle 1 (non-dosing) and then Day 1 of Cycles 2,4,6 and Cycle 10. For ''Phase 2 1L NSCLC: Utomilumab then Utomilumab + Avelumab'' reporting group: Day 1 of Cycles 2,4,6,10
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Combination A Phase 1b NSCLC: Utomilumab 500 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 20 mg + Avelumab | Combination A Phase 2 Melanoma: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCCHN: Utomilumab 100 mg + Avelumab | Combination A Phase 2 TNBC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 First Line (1L) NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 1L NSCLC: Utomilumab Then Utomilumab + Avelumab | Combination A Phase 2 1L NSCLC: Avelumab Then Utomilumab + Avelumab
Number analyzed (Participants) | 27 | 27 | 29 | 27 | 33 | 20 | 9 | 20 | 9 | 11
Nanogram per milliliter
  Cycle 1/Day1-0 Hour: number analyzed (Participants) | 27 | 26 | 29 | 27 | 33 | 20 | 9 | 20 | 0 | 11
  Cycle 1/Day1-0 Hour | 9.510 (NA) — Only 1 observation was equal or above lower limit of quantification (LLoQ). Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. | 5.532 (540) | 16.24 (19873078) | 64.96 (162) | 93.02 (190) | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | 9.440 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. | 3.082 (80) |  | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated.
  Cycle 1/Day15-0 Hour: number analyzed (Participants) | 23 | 24 | 28 | 26 | 29 | 19 | 8 | 17 | 0 | 11
  Cycle 1/Day15-0 Hour | 22.13 (106) | 17.85 (135) | 19.92 (102) | 22.02 (138) | 23.03 (74) | 25.53 (38) | 18.37 (53) | 13.15 (45) |  | 9.781 (84)
  Cycle 2/Day1-0 Hour: number analyzed (Participants) | 22 | 22 | 22 | 24 | 29 | 17 | 5 | 17 | 9 | 10
  Cycle 2/Day1-0 Hour | 23.14 (84) | 20.69 (115) | 22.67 (105) | 25.45 (224) | 23.35 (77) | 27.94 (43) | 21.61 (76) | 12.52 (80) | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | 10.96 (110)
  Cycle 4/Day1-0 Hour: number analyzed (Participants) | 14 | 8 | 11 | 10 | 15 | 9 | 3 | 6 | 8 | 6
  Cycle 4/Day1-0 Hour | 18.79 (132) | 21.53 (103) | 32.46 (74) | 49.20 (259) | 23.30 (59) | 26.82 (55) | 20.21 (86) | 26.50 (85) | 10.52 (140) | 15.38 (81)
  Cycle 6/Day1-0 Hour: number analyzed (Participants) | 10 | 4 | 6 | 5 | 11 | 7 | 2 | 5 | 6 | 6
  Cycle 6/Day1-0 Hour | 24.80 (52) | 27.33 (99) | 33.45 (40) | 59.47 (105) | 24.28 (65) | 26.17 (57) | 20.66 (9) | 27.62 (73) | 22.16 (43) | 21.05 (45)
  Cycle 10/Day1-0 Hour: number analyzed (Participants) | 7 | 3 | 4 | 4 | 5 | 3 | 0 | 3 | 2 | 4
  Cycle 10/Day1-0 Hour | 27.56 (46) | 26.87 (100) | 40.42 (66) | 39.89 (24) | 34.09 (52) | 25.31 (101) |  | 34.90 (47) | 19.04 (117) | 19.41 (24)

32. Secondary Outcome: Pre-Dose Observed Plasma Concentration (Ctrough) of Utomilumab in Combination A
Description: Ctrough is steady-state pre-dose concentration.
Time Frame: Pre-dose on Day 1 of Cycles 1,3,5,8, and Cycle 12; Day 15 of Cycle 1 (non-dosing). For ''Phase 2 1L NSCLC: Avelumab then Utomilumab + Avelumab'' reporting group: Day 1 of Cycles 3,5,8 and 12
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Combination A Phase 1b NSCLC: Utomilumab 500 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 20 mg + Avelumab | Combination A Phase 2 Melanoma: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCCHN: Utomilumab 100 mg + Avelumab | Combination A Phase 2 TNBC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 First Line (1L) NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 1L NSCLC: Utomilumab Then Utomilumab + Avelumab | Combination A Phase 2 1L NSCLC: Avelumab Then Utomilumab + Avelumab
Number analyzed (Participants) | 28 | 27 | 29 | 28 | 33 | 21 | 10 | 20 | 10 | 8
Nanogram per milliliter
  Cycle 1/Day1-0 Hour: number analyzed (Participants) | 28 | 27 | 29 | 28 | 33 | 21 | 10 | 20 | 10 | 0
  Cycle 1/Day1-0 Hour | 619.0 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | 1430 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. | 931.0 (NA) — Only 1 observation was equal or above lower limit of quantification (LLoQ). Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. | 24400 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. | 20500 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. |
  Cycle 1/Day15-0 Hour: number analyzed (Participants) | 26 | 22 | 29 | 26 | 32 | 21 | 8 | 18 | 9 | 0
  Cycle 1/Day15-0 Hour | 2723 (28) | 1536 (26) | 779.3 (25) | 1443 (20) | 1688 (23) | 2323 (30) | 2509 (28) | 2529 (49) | 4283 (42) |
  Cycle 3/Day1-0 Hour: number analyzed (Participants) | 17 | 12 | 21 | 14 | 18 | 10 | 3 | 10 | 8 | 8
  Cycle 3/Day1-0 Hour | 2114 (30) | 982.3 (29) | 743.2 (26) | 1627 (145) | 1547 (72) | 1351 (38) | 693.5 (29) | 1114 (38) | 928.0 (69) | 780.4 (48)
  Cycle 5/Day1-0 Hour: number analyzed (Participants) | 10 | 6 | 7 | 8 | 15 | 8 | 3 | 5 | 6 | 7
  Cycle 5/Day1-0 Hour | 2259 (53) | 1059 (63) | 931.9 (97) | 1281 (33) | 1366 (37) | 1417 (25) | 855.1 (14) | 1046 (30) | 906.7 (67) | 671.9 (38)
  Cycle 8/Day1-0 Hour: number analyzed (Participants) | 7 | 5 | 4 | 5 | 6 | 5 | 2 | 2 | 6 | 6
  Cycle 8/Day1-0 Hour | 1840 (54) | 1726 (21) | 839.9 (38) | 1747 (19) | 2300 (138) | 1196 (29) | 1030 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. | 1070 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. | 669.0 (27) | 851.8 (30)
  Cycle 12/Day1-0 Hour: number analyzed (Participants) | 6 | 3 | 4 | 5 | 2 | 3 | 0 | 1 | 3 | 3
  Cycle 12/Day1-0 Hour | 1814 (52) | 1171 (24) | 690.2 (35) | 1172 (39) | 610.0 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. | 1359 (5) |  | NA (NA) — There were <=2 participants, and no observation was equal or above LLoQ . Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | 655.4 (64) | 653.9 (23)

33. Secondary Outcome: Pre-Dose Observed Plasma Concentration (Ctrough) of Avelumab and PF-04518600 in Combination B
Description: Ctrough is steady-state pre-dose concentration.
Time Frame: Pre-dose on Days 1 and 15 of Cycle 1 (non-dosing); Day 1 of Cycles 2, 4, 6 and Cycle 10
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Combination B Phase 1b: PF-04518600 0.3 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 1.0 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 3.0 mg/kg + Avelumab | Combination B Phase 2 NSCLC: PF-04518600 0.3 mg/kg + Avelumab | Combination B Phase 2 SCCHN: PF-04518600 0.3 mg/kg + Avelumab
Number analyzed (Participants) | 12 | 12 | 8 | 14 | 25
Nanogram per milliliter
  Avelumab Cycle 1/Day1-0 Hour | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | 228.0 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated.
  Avelumab Cycle 1/Day15-0 Hour: number analyzed (Participants) | 10 | 11 | 6 | 13 | 22
  Avelumab Cycle 1/Day15-0 Hour | 19.05 (69) | 16.83 (63) | 19.88 (50) | 21.72 (54) | 17.00 (63)
  Avelumab Cycle 2/Day1-0 Hour: number analyzed (Participants) | 10 | 8 | 6 | 12 | 18
  Avelumab Cycle 2/Day1-0 Hour | 21.10 (84) | 21.27 (47) | 22.04 (70) | 25.32 (59) | 18.77 (92)
  Avelumab Cycle 4/Day1-0 Hour: number analyzed (Participants) | 2 | 2 | 2 | 10 | 13
  Avelumab Cycle 4/Day1-0 Hour | 15.72 (179) | 21.16 (13) | 22.37 (91) | 22.69 (46) | 17.95 (90)
  Avelumab Cycle 6/Day1-0 Hour: number analyzed (Participants) | 0 | 1 | 0 | 5 | 6
  Avelumab Cycle 6/Day1-0 Hour |  | 16.00 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. |  | 29.83 (34) | 25.82 (37)
  Avelumab Cycle 10/Day1-0 Hour: number analyzed (Participants) | 0 | 0 | 0 | 1 | 3
  Avelumab Cycle 10/Day1-0 Hour |  |  |  | 26.30 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. | 23.70 (24)
  PF-04518600 Cycle 1/Day1-0 Hour: number analyzed (Participants) | 12 | 12 | 8 | 13 | 25
  PF-04518600 Cycle 1/Day1-0 Hour | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | 5750 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. | 23.10 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated.
  PF-04518600 Cycle 1/Day15-0 Hour: number analyzed (Participants) | 10 | 11 | 6 | 13 | 22
  PF-04518600 Cycle 1/Day15-0 Hour | 1497 (55) | 6234 (50) | 25320 (29) | 1758 (59) | 1702 (50)
  PF-04518600 Cycle 2/Day1-0 Hour: number analyzed (Participants) | 11 | 8 | 7 | 13 | 23
  PF-04518600 Cycle 2/Day1-0 Hour | 1826 (176) | 11000 (23) | 31830 (99) | 2928 (39) | 2327 (58)
  PF-04518600 Cycle 4/Day1-0 Hour: number analyzed (Participants) | 3 | 0 | 3 | 10 | 13
  PF-04518600 Cycle 4/Day1-0 Hour | 2324 (235) |  | 79790 (28) | 4799 (47) | 5129 (43)
  PF-04518600 Cycle 6/Day1-0 Hour: number analyzed (Participants) | 0 | 1 | 0 | 6 | 6
  PF-04518600 Cycle 6/Day1-0 Hour |  | 17200 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. |  | 6577 (37) | 6508 (23)
  PF-04518600 Cycle 10/Day1-0 Hour: number analyzed (Participants) | 0 | 0 | 0 | 2 | 4
  PF-04518600 Cycle 10/Day1-0 Hour |  |  |  | 8097 (59) | 5484 (16)

34. Secondary Outcome: Pre-Dose Observed Plasma Concentration (Ctrough) of Avelumab and PD 0360324 in Combination C
Description: Ctrough is steady-state pre-dose concentration.
Time Frame: Pre-dose on Days 1 and 15 of Cycle 1 (non-dosing); Day 1 of Cycles 2, 4, 6 and Cycle 10
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Combination C Phase 1b: PD 0360324 50 mg + Avelumab | Combination C Phase 1b: PD 0360324 100 mg + Avelumab | Combination C Phase 1b: PD 0360324 150 mg + Avelumab
Number analyzed (Participants) | 10 | 8 | 6
Nanogram per milliliter
  Avelumab Cycle 1/Day1-0 Hour | 0.2090 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated.
  Avelumab Cycle 1/Day15-0 Hour: number analyzed (Participants) | 9 | 8 | 6
  Avelumab Cycle 1/Day15-0 Hour | 20.45 (39) | 32.34 (40) | 22.53 (63)
  Avelumab Cycle 2/Day1-0 Hour: number analyzed (Participants) | 8 | 6 | 5
  Avelumab Cycle 2/Day1-0 Hour | 16.35 (136) | 31.44 (98) | 15.94 (237)
  Avelumab Cycle 4/Day1-0 Hour: number analyzed (Participants) | 2 | 2 | 5
  Avelumab Cycle 4/Day1-0 Hour | 15.50 (23) | 57.13 (80) | 36.04 (37)
  Avelumab Cycle 6/Day1-0 Hour: number analyzed (Participants) | 2 | 1 | 2
  Avelumab Cycle 6/Day1-0 Hour | 26.38 (24) | 77.20 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. | 33.23 (15)
  Avelumab Cycle 10/Day1-0 Hour: number analyzed (Participants) | 0 | 1 | 2
  Avelumab Cycle 10/Day1-0 Hour |  | 46.90 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. | 27.09 (4)
  PD 0360324 Cycle 1/Day1-0 Hour: number analyzed (Participants) | 10 | 7 | 6
  PD 0360324 Cycle 1/Day1-0 Hour | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated.
  PD 0360324 Cycle 1/Day15-0 Hour: number analyzed (Participants) | 9 | 6 | 6
  PD 0360324 Cycle 1/Day15-0 Hour | 126.2 (20) | 390.9 (94) | 583.1 (101)
  PD 0360324 Cycle 2/Day1-0 Hour: number analyzed (Participants) | 8 | 6 | 5
  PD 0360324 Cycle 2/Day1-0 Hour | 137.7 (46) | 360.4 (110) | 2987 (105)
  PD 0360324 Cycle 4/Day1-0 Hour: number analyzed (Participants) | 2 | 2 | 5
  PD 0360324 Cycle 4/Day1-0 Hour | NA (NA) — There were <=2 participants, and no observation was equal or above LLoQ . Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | 447.2 (62) | 1397 (190)
  PD 0360324 Cycle 6/Day1-0 Hour: number analyzed (Participants) | 2 | 2 | 3
  PD 0360324 Cycle 6/Day1-0 Hour | 134.0 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. | 654.0 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. | 312.1 (128)
  PD 0360324 Cycle 10/Day1-0 Hour: number analyzed (Participants) | 0 | 1 | 1
  PD 0360324 Cycle 10/Day1-0 Hour |  | 115.0 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. | 169.0 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated.

35. Secondary Outcome: Pre-Dose Observed Plasma Concentration (Ctrough) of Avelumab in Combination D
Description: Ctrough is steady-state pre-dose concentration.
Time Frame: Pre-dose on Day 1 of Cycle 1, 2, 4, 6 and Cycle 10; Day 15 of Cycle 1 (non-dosing)
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 1.0 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 1.0 mg/kg + Avelumab
Number analyzed (Participants) | 11 | 12 | 12 | 12 | 12 | 11
Nanogram per milliliter
  Cycle 1/Day1-0 Hour | 6.200 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated.
  Cycle 1/Day15-0 Hour: number analyzed (Participants) | 11 | 11 | 12 | 8 | 12 | 7
  Cycle 1/Day15-0 Hour | 17.61 (54) | 13.22 (35) | 13.48 (38) | 17.52 (16) | 14.42 (78) | 9.445 (102)
  Cycle 2/Day1-0 Hour: number analyzed (Participants) | 11 | 10 | 11 | 7 | 10 | 7
  Cycle 2/Day1-0 Hour | 16.04 (116) | 11.04 (178) | 17.23 (31) | 11.93 (95) | 22.29 (32) | 13.19 (94)
  Cycle 4/Day1-0 Hour: number analyzed (Participants) | 5 | 5 | 6 | 3 | 7 | 3
  Cycle 4/Day1-0 Hour | 26.76 (69) | 31.10 (54) | 17.77 (27) | 24.73 (20) | 29.11 (32) | 27.00 (10)
  Cycle 6/Day1-0 Hour: number analyzed (Participants) | 4 | 5 | 4 | 2 | 3 | 2
  Cycle 6/Day1-0 Hour | 30.03 (52) | 31.36 (59) | 18.87 (17) | 27.05 (1) | 33.12 (36) | 25.26 (8)
  Cycle 10/Day1-0 Hour: number analyzed (Participants) | 3 | 4 | 4 | 2 | 2 | 2
  Cycle 10/Day1-0 Hour | 32.84 (48) | 36.98 (32) | 18.39 (26) | 35.08 (14) | 26.33 (29) | 39.35 (28)

36. Secondary Outcome: Pre-Dose Observed Plasma Concentration (Ctrough) of Utomilumab in Combination D
Description: Ctrough is steady-state pre-dose concentration.
Time Frame: Pre-dose on Day 1 of Cycle 1, 3, 5, 8 and Cycle 12; Day 15 of Cycle 1 (non-dosing)
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 1.0 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 1.0 mg/kg + Avelumab
Number analyzed (Participants) | 11 | 11 | 12 | 12 | 12 | 11
Nanogram per milliliter
  Cycle 1/Day1-0 Hour: number analyzed (Participants) | 11 | 11 | 11 | 12 | 12 | 11
  Cycle 1/Day1-0 Hour | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated.
  Cycle 1/Day15-0 Hour: number analyzed (Participants) | 9 | 10 | 12 | 9 | 12 | 9
  Cycle 1/Day15-0 Hour | 616.5 (41) | 1353 (24) | 726.4 (19) | 1649 (34) | 595.2 (23) | 1752 (16)
  Cycle 3/Day1-0 Hour: number analyzed (Participants) | 5 | 5 | 8 | 6 | 6 | 5
  Cycle 3/Day1-0 Hour | 561.0 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. | 846.0 (54) | 516.6 (31) | 602.2 (38) | 813.3 (28) | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated.
  Cycle 5/Day1-0 Hour: number analyzed (Participants) | 4 | 5 | 6 | 2 | 4 | 4
  Cycle 5/Day1-0 Hour | 712.3 (11) | 718.1 (34) | 505.0 (23) | 422.0 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. | 763.0 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated.
  Cycle 8/Day1-0 Hour: number analyzed (Participants) | 2 | 4 | 4 | 2 | 3 | 2
  Cycle 8/Day1-0 Hour | NA (NA) — There were <=2 participants, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | 730.5 (23) | 674.3 (41) | 1440 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were <=2 participants, and no observation was equal or above LLoQ . Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated.
  Cycle 12/Day1-0 Hour: number analyzed (Participants) | 2 | 4 | 3 | 2 | 1 | 0
  Cycle 12/Day1-0 Hour | 407.0 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. | 720.9 (25) | 794.2 (105) | 985.6 (81) | NA (NA) — There were <=2 participants, and no observation was equal or above LLoQ . Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. |

37. Secondary Outcome: Pre-Dose Observed Plasma Concentration (Ctrough) of PF-04518600 in Combination D
Description: Ctrough is steady-state pre-dose concentration.
Time Frame: Pre-dose on Day 1 and 15 of Cycle 1 (non-dosing); Pre-dose on Day 1 of Cycle 2, 4, 6 and Cycle 10
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 1.0 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 1.0 mg/kg + Avelumab
Number analyzed (Participants) | 11 | 11 | 12 | 11 | 12 | 11
Nanogram per milliliter
  Cycle 1/Day1-0 Hour: number analyzed (Participants) | 10 | 11 | 12 | 11 | 12 | 11
  Cycle 1/Day1-0 Hour | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated.
  Cycle 1/Day15-0 Hour: number analyzed (Participants) | 11 | 11 | 12 | 8 | 12 | 9
  Cycle 1/Day15-0 Hour | 320.2 (86) | 144.2 (128) | 1342 (50) | 1529 (31) | 6388 (22) | 5466 (30)
  Cycle 2/Day1-0 Hour: number analyzed (Participants) | 11 | 11 | 11 | 7 | 10 | 7
  Cycle 2/Day1-0 Hour | 426.0 (48) | 192.6 (168) | 1823 (121) | 2164 (31) | 11470 (19) | 8241 (86)
  Cycle 4/Day1-0 Hour: number analyzed (Participants) | 5 | 5 | 6 | 3 | 7 | 3
  Cycle 4/Day1-0 Hour | 891.8 (60) | 656.8 (101) | 4524 (32) | 3506 (38) | 24010 (16) | 21500 (12)
  Cycle 6/Day1-0 Hour: number analyzed (Participants) | 4 | 5 | 4 | 2 | 4 | 3
  Cycle 6/Day1-0 Hour | 1033 (84) | 793.4 (110) | 6712 (22) | 3971 (17) | 21990 (56) | 20230 (18)
  Cycle 10/Day1-0 Hour: number analyzed (Participants) | 3 | 4 | 4 | 2 | 2 | 2
  Cycle 10/Day1-0 Hour | 1444 (25) | 829.8 (181) | 6900 (65) | 4834 (76) | 24880 (19) | 22620 (30)

38. Secondary Outcome: Pre-Dose Observed Plasma Concentration (Ctrough) of Avelumab in Combination F
Description: Ctrough is steady-state pre-dose concentration.
Time Frame: Pre-dose on Day 1 and 15 of Cycle 1 (non-dosing); Pre-dose on Day 1 of Cycle 2, 4, 6 and Cycle 10
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Combination F Phase 1b SCCHN: CMP-001 10 mg + Avelumab | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + Utomilumab 100 mg | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + PF-04518600 0.3 mg/kg
Number analyzed (Participants) | 6 | 7 | 6
Nanogram per milliliter
  Cycle 1/Day1-0 Hour | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. | 14.30 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated.
  Cycle 1/Day15-0 Hour: number analyzed (Participants) | 5 | 5 | 6
  Cycle 1/Day15-0 Hour | 16.32 (71) | 21.26 (18) | 18.53 (68)
  Cycle 2/Day1-0 Hour: number analyzed (Participants) | 5 | 5 | 5
  Cycle 2/Day1-0 Hour | 10.97 (137) | 16.76 (122) | 18.17 (130)
  Cycle 4/Day1-0 Hour: number analyzed (Participants) | 2 | 3 | 1
  Cycle 4/Day1-0 Hour | 40.90 (20) | 24.36 (69) | 24.00 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated.
  Cycle 6/Day1-0 Hour: number analyzed (Participants) | 1 | 1 | 0
  Cycle 6/Day1-0 Hour | 37.00 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. | 31.90 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. |
  Cycle 10/Day1-0 Hour: number analyzed (Participants) | 1 | 1 | 0
  Cycle 10/Day1-0 Hour | 30.40 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. | 30.50 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. |

39. Secondary Outcome: Pre-Dose Observed Plasma Concentration (Ctrough) of Utomilumab in Combination F
Description: Ctrough is steady-state pre-dose concentration.
Time Frame: Pre-dose on Day 1 of Cycle 1 (non-dosing); Pre-dose on Day 1 of Cycle 2 and 4
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Combination F Phase 1b SCCHN: CMP-001 10 mg + Avelumab | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + Utomilumab 100 mg | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + PF-04518600 0.3 mg/kg
Number analyzed (Participants) | 0 | 7 | 0
Nanogram per milliliter
  Cycle 1/Day1-0 Hour |  | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated. |
  Cycle 2/Day1-0 Hour: number analyzed (Participants) | 0 | 6 | 0
  Cycle 2/Day1-0 Hour |  | 748.9 (25) |
  Cycle 4/Day1-0 Hour: number analyzed (Participants) | 0 | 3 | 0
  Cycle 4/Day1-0 Hour |  | 866.0 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated. |

40. Secondary Outcome: Pre-Dose Observed Plasma Concentration (Ctrough) of PF-04518600 in Combination F
Description: Ctrough is steady-state pre-dose concentration.
Time Frame: Pre-dose on Day 1 of Cycle 1 (non-dosing); Pre-dose on Day 1 of Cycles 2 and 4
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Combination F Phase 1b SCCHN: CMP-001 10 mg + Avelumab | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + Utomilumab 100 mg | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + PF-04518600 0.3 mg/kg
Number analyzed (Participants) | 0 | 0 | 6
Nanogram per milliliter
  Cycle 1/Day1-0 Hour |  |  | NA (NA) — There were >2 observations, and no observation was equal or above LLoQ. Therefore, both Geometric Mean and Geometric Coefficient of Variation could not be calculated.
  Cycle 2/Day1-0 Hour: number analyzed (Participants) | 0 | 0 | 5
  Cycle 2/Day1-0 Hour |  |  | 2179 (30)
  Cycle 4/Day1-0 Hour: number analyzed (Participants) | 0 | 0 | 1
  Cycle 4/Day1-0 Hour |  |  | 3610 (NA) — Only 1 observation was equal or above LLoQ. Only Geometric Mean was reported, and Geometric Coefficient of Variation could not be calculated.

41. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibody (ADA) Against Avelumab For Combination A
Description: ADA ever-positive was defined as at least one positive ADA result at any time point.
Time Frame: Pre-dose on Day 1 of Cycle 1, 2, 4, 6, 10. For ''Phase 2 1L NSCLC: Utomilumab then Utomilumab + Avelumab'' reporting group: Day 1 of Cycle 2, 4, 6, 10
Population: The analysis population was a subset of the safety analysis set (all participants who received at least one dose of study drug) and included participants who had at least one ADA sample collected for avelumab. Here, "Number of participants analyzed'' signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Combination A Phase 1b/2 Utomilumab 100 mg + Avelumab: During Phase 1b/2 participants with NSCLC, Melanoma, SCCHN, TNBC and SCLC received utomilumab 100 mg IV Q4W with 10 mg/kg of avelumab administered IV Q2W for 2 cycles, where each cycle was of 4 weeks.
Arm/Group | Combination A Phase 1b NSCLC: Utomilumab 500 mg + Avelumab | Combination A Phase 1b/2 Utomilumab 100 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 20 mg + Avelumab | Combination A Phase 2 1L NSCLC: Utomilumab Then Utomilumab + Avelumab | Combination A Phase 2 1L NSCLC: Avelumab Then Utomilumab + Avelumab
Number analyzed (Participants) | 29 | 141 | 29 | 11 | 11
Participants | 3 | 13 | 2 | 1 | 0

42. Secondary Outcome: Number of Participants With Positive ADA Levels Against Utomilumab For Combination A
Description: ADA ever-positive was defined as at least one positive ADA result at any time point.
Time Frame: Pre-dose on Day 1 of Cycle 1, 3, 5, 8, 12. For ''Phase 2 1L NSCLC: Avelumab then Utomilumab + Avelumab'' reporting group: Day 1 of Cycle 3, 5, 8, 12
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Arm/Group | Combination A Phase 1b NSCLC: Utomilumab 500 mg + Avelumab | Combination A Phase 1b/2 Utomilumab 100 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 20 mg + Avelumab | Combination A Phase 2 1L NSCLC: Utomilumab Then Utomilumab + Avelumab | Combination A Phase 2 1L NSCLC: Avelumab Then Utomilumab + Avelumab
Number analyzed (Participants) | 29 | 141 | 29 | 10 | 9
Participants | 6 | 51 | 16 | 7 | 6

43. Secondary Outcome: Number of Participants With Positive ADA Levels For Combination B
Description: ADA ever-positive was defined as at least one positive ADA result at any time point.
Time Frame: Pre-dose on Day 1 of Cycle 1, 2, 4, 6, and 10
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Groups:
- Combination B Phase 1b/2 PF-04518600 + Avelumab: During Phase 1b participants received PF-04518600 0.3 mg/kg and in phase 2 participants with NSCLC and SCCHN received PF-04518600 3.0 mg/kg IV Q2W with 10 mg/kg of avelumab administered IV Q2W.
Arm/Group | Combination B Phase 1b/2 PF-04518600 + Avelumab | Combination B Phase 1b: PF-04518600 1.0 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 3.0 mg/kg + Avelumab
Number analyzed (Participants) | 51 | 12 | 8
Participants
  ADA ever-positive -Avelumab | 2 | 0 | 0
  ADA ever-positive - PF-04518600 | 19 | 2 | 1

44. Secondary Outcome: Number of Participants With Positive ADA Levels For Combination C
Description: ADA ever-positive was defined as at least one positive ADA result at any time point.
Time Frame: Pre-dose on Day 1 of Cycle 1, 2, 4, 6, and 10
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Arm/Group | Combination C Phase 1b: PD 0360324 50 mg + Avelumab | Combination C Phase 1b: PD 0360324 100 mg + Avelumab | Combination C Phase 1b: PD 0360324 150 mg + Avelumab
Number analyzed (Participants) | 10 | 8 | 6
Participants
  ADA ever-positive -Avelumab | 1 | 0 | 0
  ADA ever-positive -PD 0360324 | 0 | 5 | 5

45. Secondary Outcome: Number of Participants With Positive ADA Levels Against Avelumab and PF-04518600 For Combination D
Description: ADA ever-positive was defined as at least one positive ADA result at any time point.
Time Frame: Pre-dose on Day 1 of Cycle 1, 2, 4, 6, and 10
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Arm/Group | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 1.0 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 1.0 mg/kg + Avelumab
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 11
Participants
  ADA ever-positive -Avelumab | 1 | 1 | 0 | 0 | 0 | 2
  ADA ever-positive -PF-04518600 | 5 | 7 | 6 | 2 | 3 | 1

46. Secondary Outcome: Number of Participants With Positive ADA Levels Against Utomilumab For Combination D
Description: ADA ever-positive was defined as at least one positive ADA result at any time point.
Time Frame: Pre-dose on Day 1 of Cycle 1, 3, 5, 8, 12
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Arm/Group | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 1.0 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 1.0 mg/kg + Avelumab
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 11
Participants | 3 | 4 | 7 | 5 | 5 | 5

47. Secondary Outcome: Number of Participants With Positive ADA Levels Against Avelumab and PF-04518600 For Combination F
Description: ADA ever-positive was defined as at least one positive ADA result at any time point.
Time Frame: Pre-dose on Day 1 of Cycle 1, 2, 4, 6, and 10
Population: Analysis population was subset of safety analysis set (participants who received at least one dose of study drug) and included participants who had at least one ADA sample collected for avelumab. There was no evaluable participant for PF-04518600 ADA for arms "Phase 1b SCCHN CMP-001 10 mg + Avelumab" and "Phase 1b SCCHN CMP-001 10 mg then Avelumab + Utomilumab 100 mg." Here, "Number of participants analyzed'' signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination F Phase 1b SCCHN: CMP-001 10 mg + Avelumab | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + Utomilumab 100 mg | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + PF-04518600 0.3 mg/kg
Number analyzed (Participants) | 6 | 7 | 7
Participants
  ADA ever-positive -Avelumab | 0 | 3 | 0
  ADA ever-positive - PF-04518600: number analyzed (Participants) | 0 | 0 | 7
  ADA ever-positive - PF-04518600 |  |  | 2

48. Secondary Outcome: Number of Participants With Positive ADA Levels Against Utomilumab For Combination F
Description: ADA ever-positive was defined as at least one positive ADA result at any time point.
Time Frame: Pre-dose on Day 1 of Cycle 1, 2, 4, 6, and 10
Population: Analysis population was subset of safety analysis set (participants who received at least one dose of study drug) and included participants who had at least one ADA sample collected for avelumab. There was no evaluable participant for PF-04518600 ADA for arms "Phase 1b SCCHN CMP-001 10 mg + Avelumab" and "Phase 1b SCCHN CMP-001 10 mg then Avelumab + PF-04518600 0.3 mg/kg." Here, "Number of participants analyzed'' signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination F Phase 1b SCCHN: CMP-001 10 mg + Avelumab | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + Utomilumab 100 mg | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + PF-04518600 0.3 mg/kg
Number analyzed (Participants) | 0 | 7 | 0
Participants | 0 | 5 | 0

49. Secondary Outcome: Time to Tumor Response (TTR) for Combination A
Description: TTR was defined, for participants with an objective response (confirmed CR or PR), as the time from the start date (the date of first dose of treatment) to the first documentation of objective response (CR or PR) which was subsequently confirmed. Per RECIST v1.1: CR: disappearance of all non-nodal target lesions and of all non-target lesions. In addition, any pathological lymph nodes assigned as target lesions/ non-target lesions must have a reduction in short axis to <10 mm. PR: at least a 30% decrease in sum of diameter of all target lesions, taking as reference baseline sum of diameters.
Time Frame: From first dose of study drug until first documentation of CR or PR (maximum up to 7.3 years)
Population: Analysis population included all participants who received at least one dose of study drug and who had confirmed CR or PR. Participants were classified according to study treatment actually received. If participant received more than one treatment, participant was classified according to first treatment received. Here 'number of participants analyzed' signifies participants evaluable for this outcome measure with at least 1 confirmed complete response or partial response.
Measure: Median (Full Range); unit: Months
Arm/Group | Combination A Phase 1b NSCLC: Utomilumab 500 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 20 mg + Avelumab | Combination A Phase 2 Melanoma: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCCHN: Utomilumab 100 mg + Avelumab | Combination A Phase 2 TNBC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 First Line (1L) NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 1L NSCLC: Utomilumab Then Utomilumab + Avelumab | Combination A Phase 2 1L NSCLC: Avelumab Then Utomilumab + Avelumab
Number analyzed (Participants) | 1 | 0 | 3 | 3 | 3 | 3 | 1 | 1 | 6 | 2
Months | 3.6 [3.6 to 3.6] |  | 1.9 [1.7 to 11.3] | 1.9 [1.8 to 7.4] | 1.8 [1.5 to 3.5] | 1.7 [1.6 to 1.7] | 1.7 [1.7 to 1.7] | 1.6 [1.6 to 1.6] | 3.7 [1.8 to 7.4] | 2.7 [1.6 to 3.7]

50. Secondary Outcome: TTR for Combination B
Description: as for outcome 49
Time Frame: From first dose of study drug until first documentation of CR or PR (maximum up to 7.3 years)
Population: as for outcome 49
Measure: Median (Full Range); unit: Months
Arm/Group | Combination B Phase 1b: PF-04518600 0.3 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 1.0 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 3.0 mg/kg + Avelumab | Combination B Phase 2 NSCLC: PF-04518600 0.3 mg/kg + Avelumab | Combination B Phase 2 SCCHN: PF-04518600 0.3 mg/kg + Avelumab
Number analyzed (Participants) | 0 | 0 | 0 | 2 | 2
Months |  |  |  | 2.8 [1.9 to 3.7] | 3.6 [1.7 to 5.6]

51. Secondary Outcome: TTR for Combination C
Description: as for outcome 49
Time Frame: From first dose of study drug until first documentation of CR or PR (maximum up to 7.3 years)
Population: as for outcome 49
Measure: Median (Full Range); unit: Months
Arm/Group | Combination C Phase 1b: PD 0360324 50 mg + Avelumab | Combination C Phase 1b: PD 0360324 100 mg + Avelumab | Combination C Phase 1b: PD 0360324 150 mg + Avelumab
Number analyzed (Participants) | 1 | 2 | 1
Months | 4.0 [4.0 to 4.0] | 2.8 [2.2 to 3.5] | 9.4 [9.4 to 9.4]

52. Secondary Outcome: TTR for Combination D
Description: as for outcome 49
Time Frame: From first dose of study drug until first documentation of CR or PR (maximum up to 7.3 years)
Population: as for outcome 49
Measure: Median (Full Range); unit: Months
Arm/Group | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 1.0 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 1.0 mg/kg + Avelumab
Number analyzed (Participants) | 1 | 4 | 3 | 1 | 1 | 2
Months | 3.7 [3.7 to 3.7] | 1.7 [1.7 to 3.7] | 1.6 [1.6 to 1.7] | 1.8 [1.8 to 1.8] | 1.8 [1.8 to 1.8] | 2.8 [1.9 to 3.7]

53. Secondary Outcome: TTR for Combination F
Description: as for outcome 49
Time Frame: From first dose of study drug until first documentation of CR or PR (maximum up to 7.3 years)
Population: as for outcome 49
Measure: Median (Full Range); unit: Months
Arm/Group | Combination F Phase 1b SCCHN: CMP-001 10 mg + Avelumab | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + Utomilumab 100 mg | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + PF-04518600 0.3 mg/kg
Number analyzed (Participants) | 0 | 1 | 0
Months |  | 4.4 [4.4 to 4.4] |

54. Secondary Outcome: Duration of Response (DR) for Combination A
Description: DR as assessed by investigator according to RECIST v1.1, was defined as the time from date of first documentation of objective response (CR or PR) to date of PD or death due to any cause, or data censoring date, whichever occurred first. CR: disappearance of all target and non-target lesions, and sustained for at least 4 weeks. Any pathological lymph nodes (target or non-target) reduced in short axis to <10 mm. PR: >= 30% decrease in sum of diameter of target lesions taking as reference baseline sum diameters. PD: at least a 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study treatment, with absolute increase of at least 5 mm or appearance of >=1 new lesions. DR data was censored on the date of last adequate tumor assessment for participants without an event (CR, PR, PD or death), for participants who start new anti-cancer treatment prior to DR assessment, for participants with DR assessment after >=2 missing tumor assessments.
Time Frame: From first documentation of CR or PR until first documentation of tumor progression or death due to any cause or data censoring date, whichever occurred first (maximum up to 7.3 years)
Population: Full analysis set includes all randomized participants for Cohorts A1, A2, A3, A9, and A10 and all enrolled participants for Cohorts A4, A5, A6, A7, and A8 who received at least 1 dose of study drug. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Months
Arm/Group | Combination A Phase 1b NSCLC: Utomilumab 500 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 20 mg + Avelumab | Combination A Phase 2 Melanoma: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCCHN: Utomilumab 100 mg + Avelumab | Combination A Phase 2 TNBC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 First Line (1L) NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 1L NSCLC: Utomilumab Then Utomilumab + Avelumab | Combination A Phase 2 1L NSCLC: Avelumab Then Utomilumab + Avelumab
Number analyzed (Participants) | 1 | 0 | 3 | 3 | 3 | 3 | 1 | 1 | 6 | 2
Months | 12.5 [12.5 to 12.5] |  | 27.4 [20.9 to 33.9] | 52.9 [7.9 to 53.2] | 15.8 [5.7 to 29.5] | 28.5 [3.8 to 29.7] | 3.7 [3.7 to 3.7] | 4.9 [4.9 to 4.9] | 8.1 [2.5 to 43.1] | 24.8 [5.6 to 44.0]

55. Secondary Outcome: DR for Combination B
Description: as for outcome 54
Time Frame: as for outcome 54
Population: Full analysis set included all enrolled participants who received at least one dose of study drug. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Months
Arm/Group | Combination B Phase 1b: PF-04518600 0.3 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 1.0 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 3.0 mg/kg + Avelumab | Combination B Phase 2 NSCLC: PF-04518600 0.3 mg/kg + Avelumab | Combination B Phase 2 SCCHN: PF-04518600 0.3 mg/kg + Avelumab
Number analyzed (Participants) | 0 | 0 | 0 | 2 | 2
Months |  |  |  | 5.6 [3.7 to 7.4] | 23.5 [20.9 to 26.0]

56. Secondary Outcome: DR for Combination C
Description: as for outcome 54
Time Frame: as for outcome 54
Population: as for outcome 55
Measure: Median (Full Range); unit: Months
Arm/Group | Combination C Phase 1b: PD 0360324 50 mg + Avelumab | Combination C Phase 1b: PD 0360324 100 mg + Avelumab | Combination C Phase 1b: PD 0360324 150 mg + Avelumab
Number analyzed (Participants) | 1 | 2 | 1
Months | 7.1 [7.1 to 7.1] | 7.1 [5.6 to 8.6] | 13.1 [13.1 to 13.1]

57. Secondary Outcome: DR for Combination D
Description: as for outcome 54
Time Frame: as for outcome 54
Population: as for outcome 55
Measure: Median (Full Range); unit: Months
Arm/Group | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 1.0 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 1.0 mg/kg + Avelumab
Number analyzed (Participants) | 1 | 4 | 3 | 1 | 1 | 2
Months | 5.5 [5.5 to 5.5] | 28.5 [17.5 to 49.0] | 22.1 [17.8 to 35.3] | 38.6 [38.6 to 38.6] | 26.3 [26.3 to 26.3] | 7.4 [5.6 to 9.3]

58. Secondary Outcome: DR for Combination F
Description: as for outcome 54
Time Frame: as for outcome 54
Population: Full analysis set included all randomized participants. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Months
Arm/Group | Combination F Phase 1b SCCHN: CMP-001 10 mg + Avelumab | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + Utomilumab 100 mg | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + PF-04518600 0.3 mg/kg
Number analyzed (Participants) | 0 | 1 | 0
Months |  | 18.7 [18.7 to 18.7] |

59. Secondary Outcome: Progression-free Survival (PFS) for Combination A
Description: PFS as assessed by investigator per RECIST v1.1, was defined as time (in months) from date of first dose of study drug to date of first documentation of PD or death due to any cause or data censoring date, whichever occurred first. PD: >= 20% increase in sum of diameters of target lesions, taking as a reference smallest sum on study treatment (this included baseline sum if that was smallest on study treatment). The sum must also demonstrate absolute increase of >=5 mm, or appearance of >=1 new lesions. PFS was analyzed by Kaplan-Meier method. PFS data was censored on the date the last adequate tumor assessment for participants without an event (PD or death), for participants who started new anti-cancer treatment prior to PFS event, for participants with a PFS event after >=2 missing tumor assessments.
Time Frame: From first dose of study drug until first documentation of PD or death due to any cause or data censoring date, whichever occurred first (maximum up to 7.3 years)
Population: Full analysis set includes all randomized participants for Cohorts A1, A2, A3, A9, and A10 and all enrolled participants for Cohorts A4, A5, A6, A7, and A8 who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination A Phase 1b NSCLC: Utomilumab 500 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 20 mg + Avelumab | Combination A Phase 2 Melanoma: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCCHN: Utomilumab 100 mg + Avelumab | Combination A Phase 2 TNBC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 First Line (1L) NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 1L NSCLC: Utomilumab Then Utomilumab + Avelumab | Combination A Phase 2 1L NSCLC: Avelumab Then Utomilumab + Avelumab
Number analyzed (Participants) | 29 | 28 | 29 | 28 | 35 | 21 | 10 | 21 | 11 | 11
Months | 2.2 [1.8 to 5.3] | 1.8 [1.7 to 2.3] | 1.9 [1.7 to 3.7] | 1.9 [1.8 to 3.9] | 1.9 [1.8 to 3.7] | 1.8 [1.4 to 5.5] | 1.6 [0.3 to 5.4] | 1.8 [1.7 to 3.6] | 11.9 [4.2 to NA] — Upper limit of 95% CI was not estimable as there were less number of participants with an event. | 5.5 [0.7 to 43.5]

60. Secondary Outcome: PFS for Combination B
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Full analysis set included all enrolled participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination B Phase 1b: PF-04518600 0.3 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 1.0 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 3.0 mg/kg + Avelumab | Combination B Phase 2 NSCLC: PF-04518600 0.3 mg/kg + Avelumab | Combination B Phase 2 SCCHN: PF-04518600 0.3 mg/kg + Avelumab
Number analyzed (Participants) | 12 | 12 | 8 | 14 | 25
Months | 1.7 [0.7 to 1.8] | 1.8 [1.0 to 2.7] | 1.7 [0.9 to NA] — Upper limit of 95% CI was not estimable as there were less number of participants with an event. | 3.7 [1.8 to 5.6] | 1.8 [1.7 to 2.1]

61. Secondary Outcome: PFS for Combination C
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Full analysis set included all enrolled participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination C Phase 1b: PD 0360324 50 mg + Avelumab | Combination C Phase 1b: PD 0360324 100 mg + Avelumab | Combination C Phase 1b: PD 0360324 150 mg + Avelumab
Number analyzed (Participants) | 10 | 8 | 6
Months | 1.9 [0.5 to NA] — Upper limit of 95% CI was not estimable as there were less number of participants with an event. | 9.0 [1.1 to NA] — Upper limit of 95% CI was not estimable as there were less number of participants with an event. | 12.2 [1.7 to NA] — Upper limit of 95% CI was not estimable as there were less number of participants with an event.

62. Secondary Outcome: PFS for Combination D
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Full analysis set included all enrolled participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 1.0 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 1.0 mg/kg + Avelumab
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 11
Months | 1.8 [1.1 to 9.2] | 1.8 [1.3 to NA] — Upper limit of 95% CI was not estimable as there were less number of participants with an event. | 3.7 [1.0 to 23.8] | 1.8 [1.2 to NA] — Upper limit of 95% CI was not estimable as there were less number of participants with an event. | 1.8 [1.4 to 3.1] | 1.8 [0.6 to 1.9]

63. Secondary Outcome: PFS for Combination F
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Full analysis set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination F Phase 1b SCCHN: CMP-001 10 mg + Avelumab | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + Utomilumab 100 mg | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + PF-04518600 0.3 mg/kg
Number analyzed (Participants) | 6 | 7 | 7
Months | 2.3 [1.7 to NA] — Upper limit of 95% CI was not estimable as there were less number of participants with an event. | 1.9 [1.7 to NA] — Upper limit of 95% CI was not estimable as there were less number of participants with an event. | 1.8 [1.3 to 3.6]

64. Secondary Outcome: Overall Survival (OS) for Combination A
Description: OS was defined as the time (in months) from the date of first dose of study drug to the date of death due to any cause or data censoring date, whichever occurred first. Participants last known to be alive were censored at the date of last contact. OS was analyzed by Kaplan-Meier method.
Time Frame: From first dose of study drug to date of death from any cause or data censoring date, whichever occurred first (maximum up to 7.3 years)
Population: as for outcome 59
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination A Phase 1b NSCLC: Utomilumab 500 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 20 mg + Avelumab | Combination A Phase 2 Melanoma: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCCHN: Utomilumab 100 mg + Avelumab | Combination A Phase 2 TNBC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 First Line (1L) NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 1L NSCLC: Utomilumab Then Utomilumab + Avelumab | Combination A Phase 2 1L NSCLC: Avelumab Then Utomilumab + Avelumab
Number analyzed (Participants) | 29 | 28 | 29 | 28 | 35 | 21 | 10 | 21 | 11 | 11
Months | 14.5 [6.2 to 36.1] | 12.7 [3.0 to 16.1] | 14.7 [6.8 to 22.0] | 8.1 [6.4 to 15.2] | 10.7 [7.7 to 16.9] | 10.9 [4.7 to NA] — Upper limit of 95% CI was not estimable as there were less number of participants with an event. | 11.3 [0.4 to NA] — Upper limit of 95% CI was not estimable as there were less number of participants with an event. | 12.8 [6.9 to 18.9] | 29.3 [5.8 to NA] — Upper limit of 95% CI was not estimable as there were less number of participants with an event. | 22.1 [3.4 to NA] — Upper limit of 95% CI was not estimable as there were less number of participants with an event.

65. Secondary Outcome: OS for Combination B
Description: as for outcome 64
Time Frame: as for outcome 64
Population: Full analysis set included all enrolled participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination B Phase 1b: PF-04518600 0.3 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 1.0 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 3.0 mg/kg + Avelumab | Combination B Phase 2 NSCLC: PF-04518600 0.3 mg/kg + Avelumab | Combination B Phase 2 SCCHN: PF-04518600 0.3 mg/kg + Avelumab
Number analyzed (Participants) | 12 | 12 | 8 | 14 | 25
Months | 8.5 [1.6 to NA] — Upper limit of 95% CI was not estimable as there were less number of participants with an event. | 13.5 [4.0 to NA] — Upper limit of 95% CI was not estimable as there were less number of participants with an event. | 7.1 [2.4 to 20.8] | 15.9 [6.3 to NA] — Upper limit of 95% CI was not estimable as there were less number of participants with an event. | 10.7 [6.7 to 14.5]

66. Secondary Outcome: OS for Combination C
Description: as for outcome 64
Time Frame: as for outcome 64
Population: Full analysis set included all enrolled participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination C Phase 1b: PD 0360324 50 mg + Avelumab | Combination C Phase 1b: PD 0360324 100 mg + Avelumab | Combination C Phase 1b: PD 0360324 150 mg + Avelumab
Number analyzed (Participants) | 10 | 8 | 6
Months | 16.3 [0.5 to NA] — Upper limit of 95% CI was not estimable as there were less number of participants with an event. | 30.9 [1.1 to NA] — Upper limit of 95% CI was not estimable as there were less number of participants with an event. | 17.3 [6.3 to NA] — Upper limit of 95% CI was not estimable as there were less number of participants with an event.

67. Secondary Outcome: OS for Combination D
Description: as for outcome 64
Time Frame: as for outcome 64
Population: Full analysis set included all enrolled participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 1.0 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 1.0 mg/kg + Avelumab
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 11
Months | 9.4 [3.7 to 23.5] | 7.4 [1.7 to NA] — Upper limit of 95% CI was not estimable as there were less number of participants with an event. | 16.2 [5.1 to NA] — Upper limit of 95% CI was not estimable as there were less number of participants with an event. | 6.1 [1.2 to 22.5] | 8.5 [3.4 to 25.2] | 6.6 [1.8 to NA] — Upper limit of 95% CI was not estimable as there were less number of participants with an event.

68. Secondary Outcome: OS for Combination F
Description: as for outcome 64
Time Frame: as for outcome 64
Population: Full analysis set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination F Phase 1b SCCHN: CMP-001 10 mg + Avelumab | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + Utomilumab 100 mg | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + PF-04518600 0.3 mg/kg
Number analyzed (Participants) | 6 | 7 | 7
Months | 10.0 [2.2 to NA] — Upper limit of 95% CI was not estimable as there were less number of participants with an event. | 11.7 [2.0 to NA] — Upper limit of 95% CI was not estimable as there were less number of participants with an event. | 5.9 [3.0 to 7.9]

69. Secondary Outcome: Phase 1b: Percentage of Participants With Objective Response (OR) for Combination A
Description: OR as assessed by investigator per RECIST v.1.1, was defined as participants with confirmed best overall response of complete response (CR) or partial response (PR), were recorded from first dose of study drug until disease progression or death due to any cause. CR was defined as disappearance of all target and non-target lesions, and sustained for at least 4 weeks. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 mm. PR was defined as >=30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose of study drug until disease progression or death due to any cause (maximum up to 7.3 years)
Population: as for outcome 59
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Combination A Phase 1b NSCLC: Utomilumab 500 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 20 mg + Avelumab
Number analyzed (Participants) | 29 | 28 | 29
Percentage of participants | 3.4 [0.1 to 17.8] | 0 [0.0 to 12.3] | 10.3 [2.2 to 27.4]

70. Secondary Outcome: Phase 1b: Percentage of Participants With Objective Response (OR) for Combination B
Description: OR as assessed by investigator per RECIST v.1.1, was defined as participants with confirmed best overall response of CR or PR, were recorded from first dose of study drug until disease progression or death due to any cause. CR was defined as disappearance of all target and non-target lesions, and sustained for at least 4 weeks. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 mm. PR was defined as >=30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose of study drug until disease progression or death due to any cause (maximum up to 7.3 years)
Population: Full analysis set included all enrolled participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Combination B Phase 1b: PF-04518600 0.3 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 1.0 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 3.0 mg/kg + Avelumab
Number analyzed (Participants) | 12 | 12 | 8
Percentage of participants | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 36.9]

71. Secondary Outcome: Phase 1b: Percentage of Participants With Objective Response (OR) for Combination C
Description: as for outcome 70
Time Frame: From first dose of study drug until disease progression or death due to any cause (maximum up to 7.3 years)
Population: Full analysis set included all enrolled participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Combination C Phase 1b: PD 0360324 50 mg + Avelumab | Combination C Phase 1b: PD 0360324 100 mg + Avelumab | Combination C Phase 1b: PD 0360324 150 mg + Avelumab
Number analyzed (Participants) | 10 | 8 | 6
Percentage of participants | 10.0 [0.3 to 44.5] | 25.0 [3.2 to 65.1] | 16.7 [0.4 to 64.1]

72. Secondary Outcome: Phase 1b: Percentage of Participants With Objective Response (OR) for Combination D
Description: as for outcome 70
Time Frame: From first dose of study drug until disease progression or death due to any cause (maximum up to 7.3 years)
Population: Full analysis set included all enrolled participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 1.0 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 1.0 mg/kg + Avelumab
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 11
Percentage of participants | 8.3 [0.2 to 38.5] | 33.3 [9.9 to 65.1] | 25.0 [5.5 to 57.2] | 8.3 [0.2 to 38.5] | 8.3 [0.2 to 38.5] | 18.2 [2.3 to 51.8]

73. Secondary Outcome: Phase 1b: Percentage of Participants With Objective Response (OR) for Combination F
Description: as for outcome 70
Time Frame: From first dose of study drug until disease progression or death due to any cause (maximum up to 7.3 years)
Population: Full analysis set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Combination F Phase 1b SCCHN: CMP-001 10 mg + Avelumab | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + Utomilumab 100 mg | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + PF-04518600 0.3 mg/kg
Number analyzed (Participants) | 6 | 7 | 7
Percentage of participants | 0 [0.0 to 45.9] | 14.3 [0.4 to 57.9] | 0 [0.0 to 41.0]

74. Secondary Outcome: Number of Participants With Positive Programmed Death Ligand-1 (PD-L1) Biomarker Expression and Tumor Infiltrating Cluster of Differentiation 8 (CD8+) Lymphocytes at Baseline for Combination A
Description: PD-L1 protein expression is determined by using Tumor Proportion Score (TPS), which is the percentage of viable tumor cells showing partial or complete membrane staining at any intensity. The specimen is considered to have PD-L1 expression if TPS >=1% and high PD-L1 expression if TPS >= 50%. Tumor infiltrating CD8+ lymphocytes is defined as the number of CD8+ cells per unit area and the percent of counted cells. Positive is defined as >=1% and negative is defined as <1%.
Time Frame: Baseline (Day 1)
Population: The analysis population was a subset of the safety analysis set (all participants who received at least one dose of study drug) and included participants who had at least one biomarker parameter of PD-L1 and CD8+ lymphocytes from the corresponding assay sample with at least one baseline biomarker measurement. Here, ''Number Analyzed'' signifies number of participants evaluable for each specified row.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination A Phase 1b NSCLC: Utomilumab 500 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 20 mg + Avelumab | Combination A Phase 2 Melanoma: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCCHN: Utomilumab 100 mg + Avelumab | Combination A Phase 2 TNBC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 First Line (1L) NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 1L NSCLC: Utomilumab Then Utomilumab + Avelumab | Combination A Phase 2 1L NSCLC: Avelumab Then Utomilumab + Avelumab
Number analyzed (Participants) | 24 | 24 | 22 | 22 | 24 | 18 | 8 | 18 | 9 | 8
Participants
  PD-L1 | 24 | 24 | 22 | 22 | 24 | 18 | 8 | 18 | 9 | 8
  CD8+: number analyzed (Participants) | 24 | 24 | 22 | 21 | 24 | 18 | 8 | 18 | 9 | 8
  CD8+ | 24 | 24 | 22 | 21 | 24 | 18 | 8 | 18 | 9 | 8

75. Secondary Outcome: Number of Participants With Positive Programmed Death Ligand-1 (PD-L1) Biomarker Expression and Tumor Infiltrating CD8+ Lymphocytes at Baseline for Combination B
Description: PD-L1 protein expression is determined by using TPS, which is the percentage of viable tumor cells showing partial or complete membrane staining at any intensity. The specimen is considered to have PD-L1 expression if TPS >=1% and high PD-L1 expression if TPS >= 50%. Tumor infiltrating CD8+ lymphocytes is defined as the number of CD8+ cells per unit area and the percent of counted cells. Positive is defined as >=1% and negative is defined as <1%.
Time Frame: Baseline (Day 1)
Population: The analysis population was a subset of the safety analysis set (all participants who received at least one dose of study drug) and included participants who had at least one biomarker parameter of PD-L1 and CD8+ lymphocytes from the corresponding assay sample with at least one baseline biomarker measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination B Phase 1b: PF-04518600 0.3 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 1.0 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 3.0 mg/kg + Avelumab | Combination B Phase 2 NSCLC: PF-04518600 0.3 mg/kg + Avelumab | Combination B Phase 2 SCCHN: PF-04518600 0.3 mg/kg + Avelumab
Number analyzed (Participants) | 4 | 8 | 4 | 10 | 19
Participants
  PD-L1 | 4 | 8 | 4 | 10 | 19
  CD8+ | 3 | 8 | 4 | 10 | 18

76. Secondary Outcome: Number of Participants With Positive Programmed Death Ligand-1 (PD-L1) Biomarker Expression and Tumor Infiltrating CD8+ Lymphocytes at Baseline for Combination C
Description: as for outcome 75
Time Frame: Baseline (Day 1)
Population: as for outcome 75
Measure: Count of Participants; unit: Participants
Arm/Group | Combination C Phase 1b: PD 0360324 50 mg + Avelumab | Combination C Phase 1b: PD 0360324 100 mg + Avelumab | Combination C Phase 1b: PD 0360324 150 mg + Avelumab
Number analyzed (Participants) | 6 | 3 | 4
Participants
  PD-L1 | 6 | 3 | 4
  CD8+ | 6 | 3 | 4

77. Secondary Outcome: Number of Participants With Positive Programmed Death Ligand-1 (PD-L1) Biomarker Expression and Tumor Infiltrating CD8+ Lymphocytes at Baseline for Combination D
Description: as for outcome 75
Time Frame: Baseline (Day 1)
Population: as for outcome 75
Measure: Count of Participants; unit: Participants
Arm/Group | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 1.0 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 1.0 mg/kg + Avelumab
Number analyzed (Participants) | 9 | 8 | 11 | 10 | 10 | 10
Participants
  PD-L1 | 9 | 8 | 11 | 10 | 10 | 10
  CD8+ | 8 | 8 | 11 | 9 | 10 | 10

78. Secondary Outcome: Number of Participants With Positive Programmed Death Ligand-1 (PD-L1) Biomarker Expression and Tumor Infiltrating CD8+ Lymphocytes at Baseline for Combination F
Description: as for outcome 75
Time Frame: Baseline (Day 1)
Population: as for outcome 75
Measure: Count of Participants; unit: Participants
Arm/Group | Combination F Phase 1b SCCHN: CMP-001 10 mg + Avelumab | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + Utomilumab 100 mg | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + PF-04518600 0.3 mg/kg
Number analyzed (Participants) | 4 | 7 | 5
Participants
  PD-L1 | 4 | 7 | 5
  CD8+ | 4 | 7 | 5

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days post last dose (upto a maximum of 6.5 years [Combination-A], 3.5 years [Combination-B], 1.8 years [Combination-C], 4.3 years [Combination-D] and 3 years [Combination-F]). All-Cause Mortality was from randomization until death, assessed up to 7.3 years.
Description: The same event may appear as both AE and SAE. An event may be categorized as serious in 1 participant and non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study. For AE and SAE safety analysis set was analyzed. Safety analysis set includes all participants who received at least 1 dose of study drug. For All-Cause Mortality full analysis set was analyzed. Full analysis set includes all randomized participants in the study.
Arm/Group | Combination A Phase 1b NSCLC: Utomilumab 500 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 1b NSCLC: Utomilumab 20 mg + Avelumab | Combination A Phase 2 Melanoma: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCCHN: Utomilumab 100 mg + Avelumab | Combination A Phase 2 TNBC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 SCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 First Line (1L) NSCLC: Utomilumab 100 mg + Avelumab | Combination A Phase 2 1L NSCLC: Utomilumab Then Utomilumab + Avelumab | Combination A Phase 2 1L NSCLC: Avelumab Then Utomilumab + Avelumab | Combination B Phase 1b: PF-04518600 0.3 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 1.0 mg/kg + Avelumab | Combination B Phase 1b: PF-04518600 3.0 mg/kg + Avelumab | Combination B Phase 2 NSCLC: PF-04518600 0.3 mg/kg + Avelumab | Combination B Phase 2 SCCHN: PF-04518600 0.3 mg/kg + Avelumab | Combination C Phase 1b: PD 0360324 50 mg + Avelumab | Combination C Phase 1b: PD 0360324 100 mg + Avelumab | Combination C Phase 1b: PD 0360324 150 mg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.1 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.3 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 1.0 mg/kg + Avelumab | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 1.0 mg/kg + Avelumab | Combination F Phase 1b SCCHN: CMP-001 10 mg + Avelumab | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + Utomilumab 100 mg | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + PF-04518600 0.3 mg/kg
All-Cause Mortality (participants affected / at risk) | 18/29 | 19/28 | 20/29 | 19/28 | 25/35 | 12/21 | 6/10 | 14/21 | 7/11 | 6/11 | 7/12 | 6/12 | 6/8 | 8/14 | 21/25 | 5/10 | 4/8 | 4/6 | 9/12 | 7/12 | 7/12 | 8/12 | 10/12 | 7/11 | 4/6 | 5/7 | 7/7
Serious Adverse Events (participants affected / at risk) | 11/29 | 12/27 | 13/29 | 9/28 | 16/35 | 4/21 | 4/10 | 8/21 | 4/11 | 1/11 | 3/12 | 4/12 | 1/8 | 3/14 | 10/25 | 4/10 | 3/8 | 4/6 | 2/12 | 3/12 | 4/12 | 5/12 | 4/12 | 5/11 | 2/6 | 4/7 | 4/7
Other Adverse Events (participants affected / at risk) | 29/29 | 27/27 | 28/29 | 28/28 | 33/35 | 20/21 | 10/10 | 21/21 | 11/11 | 10/11 | 12/12 | 12/12 | 8/8 | 14/14 | 25/25 | 9/10 | 8/8 | 6/6 | 12/12 | 11/12 | 12/12 | 11/12 | 12/12 | 11/11 | 5/6 | 7/7 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination A Phase 1b NSCLC: Utomilumab 500 mg + Avelumab (N=29) | Combination A Phase 1b NSCLC: Utomilumab 100 mg + Avelumab (N=27) | Combination A Phase 1b NSCLC: Utomilumab 20 mg + Avelumab (N=29) | Combination A Phase 2 Melanoma: Utomilumab 100 mg + Avelumab (N=28) | Combination A Phase 2 SCCHN: Utomilumab 100 mg + Avelumab (N=35) | Combination A Phase 2 TNBC: Utomilumab 100 mg + Avelumab (N=21) | Combination A Phase 2 SCLC: Utomilumab 100 mg + Avelumab (N=10) | Combination A Phase 2 First Line (1L) NSCLC: Utomilumab 100 mg + Avelumab (N=21) | Combination A Phase 2 1L NSCLC: Utomilumab Then Utomilumab + Avelumab (N=11) | Combination A Phase 2 1L NSCLC: Avelumab Then Utomilumab + Avelumab (N=11) | Combination B Phase 1b: PF-04518600 0.3 mg/kg + Avelumab (N=12) | Combination B Phase 1b: PF-04518600 1.0 mg/kg + Avelumab (N=12) | Combination B Phase 1b: PF-04518600 3.0 mg/kg + Avelumab (N=8) | Combination B Phase 2 NSCLC: PF-04518600 0.3 mg/kg + Avelumab (N=14) | Combination B Phase 2 SCCHN: PF-04518600 0.3 mg/kg + Avelumab (N=25) | Combination C Phase 1b: PD 0360324 50 mg + Avelumab (N=10) | Combination C Phase 1b: PD 0360324 100 mg + Avelumab (N=8) | Combination C Phase 1b: PD 0360324 150 mg + Avelumab (N=6) | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.1 mg/kg + Avelumab (N=12) | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.1 mg/kg + Avelumab (N=12) | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.3 mg/kg + Avelumab (N=12) | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.3 mg/kg + Avelumab (N=12) | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 1.0 mg/kg + Avelumab (N=12) | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 1.0 mg/kg + Avelumab (N=11) | Combination F Phase 1b SCCHN: CMP-001 10 mg + Avelumab (N=6) | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + Utomilumab 100 mg (N=7) | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + PF-04518600 0.3 mg/kg (N=7)
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 2 | 4 | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungaemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Phlebitis infective (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blindness (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacunar infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral cavity fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combination A Phase 1b NSCLC: Utomilumab 500 mg + Avelumab (N=29) | Combination A Phase 1b NSCLC: Utomilumab 100 mg + Avelumab (N=27) | Combination A Phase 1b NSCLC: Utomilumab 20 mg + Avelumab (N=29) | Combination A Phase 2 Melanoma: Utomilumab 100 mg + Avelumab (N=28) | Combination A Phase 2 SCCHN: Utomilumab 100 mg + Avelumab (N=35) | Combination A Phase 2 TNBC: Utomilumab 100 mg + Avelumab (N=21) | Combination A Phase 2 SCLC: Utomilumab 100 mg + Avelumab (N=10) | Combination A Phase 2 First Line (1L) NSCLC: Utomilumab 100 mg + Avelumab (N=21) | Combination A Phase 2 1L NSCLC: Utomilumab Then Utomilumab + Avelumab (N=11) | Combination A Phase 2 1L NSCLC: Avelumab Then Utomilumab + Avelumab (N=11) | Combination B Phase 1b: PF-04518600 0.3 mg/kg + Avelumab (N=12) | Combination B Phase 1b: PF-04518600 1.0 mg/kg + Avelumab (N=12) | Combination B Phase 1b: PF-04518600 3.0 mg/kg + Avelumab (N=8) | Combination B Phase 2 NSCLC: PF-04518600 0.3 mg/kg + Avelumab (N=14) | Combination B Phase 2 SCCHN: PF-04518600 0.3 mg/kg + Avelumab (N=25) | Combination C Phase 1b: PD 0360324 50 mg + Avelumab (N=10) | Combination C Phase 1b: PD 0360324 100 mg + Avelumab (N=8) | Combination C Phase 1b: PD 0360324 150 mg + Avelumab (N=6) | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.1 mg/kg + Avelumab (N=12) | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.1 mg/kg + Avelumab (N=12) | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 0.3 mg/kg + Avelumab (N=12) | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 0.3 mg/kg + Avelumab (N=12) | Combination D Phase 1b: Utomilumab 20 mg + PF-04518600 1.0 mg/kg + Avelumab (N=12) | Combination D Phase 1b: Utomilumab 50 mg + PF-04518600 1.0 mg/kg + Avelumab (N=11) | Combination F Phase 1b SCCHN: CMP-001 10 mg + Avelumab (N=6) | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + Utomilumab 100 mg (N=7) | Combination F Phase 1b SCCHN: CMP-001 10 mg Then Avelumab + PF-04518600 0.3 mg/kg (N=7)
Anaemia (Blood and lymphatic system disorders) | 2 | 4 | 1 | 1 | 6 | 2 | 1 | 2 | 1 | 3 | 1 | 3 | 1 | 2 | 1 | 1 | 1 | 0 | 2 | 1 | 2 | 2 | 1 | 2 | 1 | 2 | 3
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial thrombosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 4 | 2 | 1 | 2 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 4 | 2 | 5 | 0 | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 1 | 0 | 2 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular discomfort (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 2 | 0 | 5 | 2 | 1 | 0 | 4 | 2 | 2 | 3 | 1 | 1 | 2 | 4 | 1 | 0 | 1 | 2 | 1 | 0 | 2 | 0 | 3 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 1 | 2 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Angular cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 4 | 4 | 8 | 8 | 6 | 3 | 2 | 5 | 3 | 1 | 3 | 4 | 1 | 2 | 5 | 1 | 2 | 1 | 3 | 4 | 2 | 0 | 1 | 0 | 0 | 5 | 2
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 5 | 6 | 5 | 7 | 4 | 2 | 6 | 3 | 2 | 2 | 1 | 4 | 6 | 4 | 2 | 1 | 2 | 5 | 2 | 4 | 2 | 3 | 2 | 3 | 4 | 1
Dry mouth (Gastrointestinal disorders) | 3 | 5 | 0 | 3 | 2 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 1 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 3 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 3 | 1 | 1 | 3 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 | 9 | 7 | 8 | 2 | 4 | 3 | 9 | 5 | 3 | 5 | 1 | 1 | 4 | 6 | 2 | 3 | 3 | 0 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 2
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal spasm (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 6 | 7 | 5 | 6 | 7 | 6 | 1 | 4 | 2 | 4 | 4 | 0 | 2 | 5 | 3 | 3 | 2 | 4 | 0 | 1 | 2 | 4 | 3 | 3 | 3 | 2 | 1
Asthenia (General disorders) | 1 | 3 | 5 | 2 | 5 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 2
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 4 | 4 | 1 | 4 | 4 | 5 | 1 | 6 | 2 | 4 | 1 | 0 | 0 | 3 | 3 | 2 | 1 | 0 | 3 | 2 | 2 | 2 | 3 | 2 | 2 | 3 | 4
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 10 | 14 | 12 | 11 | 8 | 3 | 3 | 9 | 7 | 4 | 7 | 5 | 2 | 4 | 7 | 3 | 2 | 1 | 5 | 5 | 6 | 5 | 6 | 2 | 5 | 4 | 6
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ill-defined disorder (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 1 | 2 | 2 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 2 | 2 | 4 | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Pain (General disorders) | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 3 | 3 | 4 | 3 | 5 | 4 | 2 | 2 | 1 | 2 | 0 | 2 | 0 | 3 | 1 | 1 | 1 | 1 | 1 | 2 | 2 | 1 | 0 | 2 | 2 | 2 | 2
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swelling face (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 0
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fungal foot infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lip infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lyme disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 2 | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 5 | 2 | 1 | 2 | 3 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 3 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 1 | 3 | 0 | 2 | 0 | 2 | 2 | 2 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 4 | 4 | 0 | 1 | 1 | 2 | 4 | 2 | 3 | 0 | 1 | 1 | 2 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incision site erythema (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 10 | 4 | 7 | 3 | 3 | 3 | 2 | 1 | 1 | 2 | 3 | 4 | 2 | 2 | 0 | 0 | 1 | 2 | 1 | 3 | 1 | 4 | 2 | 3 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac valve disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulseless electrical activity (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Secondary hypogonadism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Visual field defect (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Swelling of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pterygium (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tooth discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal pruritus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site related reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Necrosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug withdrawal syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Induration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hernia pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impaired healing (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Medical device site burn (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contrast media allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pilonidal disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Catheter site cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes dermatitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infected skin ulcer (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Penile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Sialoadenitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1 | 1 | 1 | 2 | 1 | 0 | 3 | 0 | 3 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 3 | 1 | 2 | 4 | 1 | 0 | 3 | 1 | 4 | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood calcium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 1 | 2 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 2 | 1 | 2 | 1 | 0 | 2 | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 1 | 2 | 3 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 1 | 4 | 1 | 5 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 1 | 1 | 6 | 3 | 1 | 0 | 1 | 1 | 3 | 0 | 1 | 1 | 2 | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 3 | 5 | 4 | 2 | 3 | 0 | 3 | 1 | 0 | 3 | 0 | 1 | 3 | 4 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 3 | 0 | 1 | 2 | 1
Weight increased (Investigations) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 3 | 9 | 2 | 5 | 4 | 6 | 6 | 2 | 3 | 0 | 2 | 3 | 5 | 6 | 3 | 3 | 1 | 1 | 1 | 1 | 3 | 3 | 3 | 1 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 3 | 4 | 5 | 2 | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 4 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1 | 4 | 3 | 5 | 3 | 3 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 0 | 2 | 1 | 0 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 3 | 0 | 1 | 2 | 1 | 2 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 3 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 4 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 4 | 4 | 3 | 3 | 4 | 1 | 5 | 4 | 4 | 2 | 3 | 1 | 3 | 3 | 0 | 2 | 1 | 1 | 4 | 3 | 1 | 3 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 3 | 3 | 5 | 4 | 7 | 0 | 4 | 3 | 5 | 2 | 1 | 0 | 2 | 2 | 1 | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 2 | 1 | 3 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 3 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 0 | 1 | 3 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 4 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 3 | 0 | 1 | 4 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 3 | 5 | 0 | 0 | 4 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 2 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 3 | 3 | 1 | 2 | 3 | 1 | 1 | 1 | 4 | 1 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 3 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 3 | 3 | 2 | 5 | 1 | 1 | 3 | 1 | 2 | 1 | 2 | 0 | 0 | 4 | 1 | 3 | 1 | 0 | 2 | 1 | 1 | 3 | 2 | 1 | 1 | 1
Dysgeusia (Nervous system disorders) | 3 | 1 | 1 | 0 | 1 | 2 | 1 | 3 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 5 | 6 | 1 | 2 | 4 | 2 | 1 | 3 | 4 | 4 | 1 | 0 | 1 | 0 | 6 | 1 | 3 | 2 | 1 | 5 | 3 | 3 | 5 | 3 | 2 | 2 | 2
Intention tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 2 | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 2 | 3 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Depression (Psychiatric disorders) | 2 | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 1 | 4 | 2 | 2 | 2 | 2 | 1 | 2 | 0 | 2 | 2 | 0 | 5 | 2 | 1 | 3 | 2 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 8 | 2 | 5 | 3 | 1 | 4 | 2 | 5 | 3 | 1 | 0 | 2 | 2 | 2 | 1 | 0 | 2 | 3 | 4 | 3 | 4 | 2 | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 8 | 2 | 7 | 4 | 4 | 4 | 5 | 5 | 3 | 1 | 1 | 7 | 5 | 3 | 2 | 2 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 0 | 2 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 2 | 2 | 0 | 0 | 0 | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 1 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 2 | 2 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymph node palpable (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amylase (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood creatine phosphokinase (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood corticotrophin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood corticotrophin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pancreatic enzymes increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Limb mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device occlusion (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysmetria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Generalised anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Central nervous system lesion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness exertional (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Superior sagittal sinus thrombosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anticipatory anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Testicular swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peyronie's disease (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngeal reflux (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 4 | 1 | 1 | 2 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 7 | 2 | 4 | 4 | 3 | 3 | 2 | 3 | 2 | 1 | 1 | 2 | 1 | 4 | 1 | 0 | 2 | 2 | 4 | 2 | 2 | 5 | 2 | 1 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 4 | 1 | 4 | 2 | 0 | 0 | 2 | 1 | 3 | 1 | 0 | 0 | 2 | 3 | 1 | 0 | 1 | 1 | 3 | 3 | 2 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 2 | 1 | 2 | 1 | 1 | 3 | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 2 | 3 | 3 | 2 | 0 | 1 | 0 | 0 | 2
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Butterfly rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail pitting (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus operation (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Hypertension (Vascular disorders) | 1 | 0 | 1 | 2 | 2 | 0 | 0 | 3 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 2 | 1 | 2 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 2 | 2
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral venous disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Scalp haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Superficial vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
For combination C and D the level of clinical activity observed in Cohorts C11 to C13 and D11 to D32 did not support development beyond Phase 1b. For combination F, the level of clinical activity did not warrant further enrolment. Therefore, Phase 2 was not planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-12-13): https://cdn.clinicaltrials.gov/large-docs/12/NCT02554812/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/12/NCT02554812/SAP_001.pdf